CLINICAL TRIAL: NCT00529373
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Assess the Safety and Efficacy of Odanacatib (MK-0822) to Reduce the Risk of Fracture in Osteoporotic Postmenopausal Women Treated With Vitamin D and Calcium
Brief Title: A Study of MK-0822 in Postmenopausal Women With Osteoporosis to Assess Fracture Risk (MK-0822-018)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-018; 2007_610; 132238 (Registry Identifier: JAPIC-CTI); 2007-002693-66 (EudraCT Number)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — odanacatib; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odanacatib (Experimental): Participants receive 50 mg of blinded odanacatib weekly over the course of the base study and first extension study (5 years total), followed by 50 mg of open-label odanacatib weekly for 5 years. Participants also receive Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) is approximately 1200 mg.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Placebo (Placebo Comparator): Participants receive blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total), followed by 50 mg of open-label odanacatib weekly for 5 years. Participants also receive Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) is approximately 1200 mg.
  Interventions: Drug: Placebo for Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: Odanacatib — 50 mg tablet orally once weekly (OW)
  Other Names: MK-0822
  Arms: Odanacatib
Drug: Placebo for Odanacatib — 50 mg tablet orally OW
  Arms: Placebo
Dietary Supplement: Vitamin D3 — 5600 IU orally OW
Dietary Supplement: Calcium carbonate — If needed. Total daily calcium intake (from both dietary and supplemental sources) will be approximately 1200 mg but not to exceed 1600 mg
  Other Names: Calcium supplements

SUMMARY:
The purpose of the event-driven base study is to determine the safety and efficacy, especially fracture risk reduction, of odanacatib in postmenopausal women diagnosed with osteoporosis. In a placebo-controlled extension of the base study, participants continued to receive the same blinded study medication for a total of up to 5 years of blinded study medication combined between the base study and the extension. After participants received 5 years of blinded study medication, they received open-label odanacatib through the end of the first extension. Participants were then invited to enroll in a second extension study in which they received open-label odanacatib for an additional 5 years. Two imaging substudies (PN032-Base/Extension and PN035) were conducted for participants in the MK-0822-018 Study. Additional safety information was collected for participants who discontinued from the base study or the blinded first extension in an observational follow-up study, MK-0822-083 (EudraCT number: 2007-002693-66) .

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (for at least 5 years) who are ≥65 years of age and have low bone mineral density
* Ambulatory (able to walk)

Exclusion Criteria:

* Must not be taking osteoporosis therapy or have a metabolic bone disorder other than osteoporosis
* Has or has had a hip fracture
* Currently participating in another drug study

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16071 (Actual)
Dates: Start 2007-09-13 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2017-02-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Bone HG, Dempster DW, Eisman JA, Greenspan SL, McClung MR, Nakamura T, Papapoulos S, Shih WJ, Rybak-Feiglin A, Santora AC, Verbruggen N, Leung AT, Lombardi A. Odanacatib for the treatment of postmenopausal osteoporosis: development history and design and participant characteristics of LOFT, the Long-Term Odanacatib Fracture Trial. Osteoporos Int. 2015 Feb;26(2):699-712. doi: 10.1007/s00198-014-2944-6. Epub 2014 Nov 29. PMID 25432773
- [Derived] Duong LT, Clark S, Pickarski M, Giezek H, Cohn D, Massaad R, Stoch SA. Effects of odanacatib on bone-turnover markers in osteoporotic postmenopausal women: a post hoc analysis of the LOFT study. Osteoporos Int. 2022 Oct;33(10):2165-2175. doi: 10.1007/s00198-022-06406-x. Epub 2022 Jun 17. PMID 35711006
- [Derived] Papapoulos S, Bone H, Cosman F, Dempster DW, McClung MR, Nakamura T, Restrepo JFM, Bouxsein ML, Cohn D, de Papp A, Massaad R, Santora A. Incidence of Hip and Subtrochanteric/Femoral Shaft Fractures in Postmenopausal Women With Osteoporosis in the Phase 3 Long-Term Odanacatib Fracture Trial. J Bone Miner Res. 2021 Jul;36(7):1225-1234. doi: 10.1002/jbmr.4284. Epub 2021 Apr 27. PMID 33724542
- [Derived] Recker R, Dempster D, Langdahl B, Giezek H, Clark S, Ellis G, de Villiers T, Valter I, Zerbini CA, Cohn D, Santora A, Duong LT. Effects of Odanacatib on Bone Structure and Quality in Postmenopausal Women With Osteoporosis: 5-Year Data From the Phase 3 Long-Term Odanacatib Fracture Trial (LOFT) and its Extension. J Bone Miner Res. 2020 Jul;35(7):1289-1299. doi: 10.1002/jbmr.3994. Epub 2020 May 5. PMID 32119749
- [Derived] McClung MR, O'Donoghue ML, Papapoulos SE, Bone H, Langdahl B, Saag KG, Reid IR, Kiel DP, Cavallari I, Bonaca MP, Wiviott SD, de Villiers T, Ling X, Lippuner K, Nakamura T, Reginster JY, Rodriguez-Portales JA, Roux C, Zanchetta J, Zerbini CAF, Park JG, Im K, Cange A, Grip LT, Heyden N, DaSilva C, Cohn D, Massaad R, Scott BB, Verbruggen N, Gurner D, Miller DL, Blair ML, Polis AB, Stoch SA, Santora A, Lombardi A, Leung AT, Kaufman KD, Sabatine MS; LOFT Investigators. Odanacatib for the treatment of postmenopausal osteoporosis: results of the LOFT multicentre, randomised, double-blind, placebo-controlled trial and LOFT Extension study. Lancet Diabetes Endocrinol. 2019 Dec;7(12):899-911. doi: 10.1016/S2213-8587(19)30346-8. Epub 2019 Oct 31. PMID 31676222

RESULTS

PARTICIPANT FLOW:
Groups:
- Odanacatib 50 mg OW: Participants received 50 mg of blinded odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for up to 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
- Placebo: Participants received blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for up to 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Period: Base Study
Arm/Group | Odanacatib 50 mg OW | Placebo
Started | 8043 | 8028
Completed | 4297 | 3960
Not Completed | 3746 | 4068
Not completed — Adverse Event | 525 | 470
Not completed — Lack of Efficacy | 16 | 75
Not completed — Lost to Follow-up | 221 | 208
Not completed — Other Protocol Specified Criteria | 19 | 20
Not completed — Physician Decision | 60 | 52
Not completed — Protocol Violation | 48 | 38
Not completed — Withdrawal by Subject | 1062 | 967
Not completed — Did not continue into Extension | 1795 | 2238
Period: First Extension Study
Arm/Group | Odanacatib 50 mg OW | Placebo
Started | 4297 | 3960
Completed | 3144 | 2309
Not Completed | 1153 | 1651
Not completed — Adverse Event | 162 | 142
Not completed — Lack of Efficacy | 65 | 427
Not completed — Lost to Follow-up | 41 | 37
Not completed — Other | 27 | 47
Not completed — Physician Decision | 50 | 45
Not completed — Protocol Violation | 16 | 13
Not completed — Withdrawal by Subject | 296 | 287
Not completed — Disposition record non-existing | 0 | 1
Not completed — Discontinued after 5 years completion | 208 | 346
Not completed — Did not cont. into 2nd Ext (verified) | 256 | 281
Not completed — Did not cont. into 2nd Ext (unknown) | 32 | 25
Period: Second Extension Study
Arm/Group | Odanacatib 50 mg OW | Placebo
Started | 3144 | 2309
Completed | 2844 | 2112
Not Completed | 300 | 197
Not completed — Adverse Event | 101 | 51
Not completed — Lack of Efficacy | 7 | 15
Not completed — Lost to Follow-up | 18 | 12
Not completed — Other | 7 | 12
Not completed — Physician Decision | 63 | 26
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 97 | 75
Not completed — Status Missing | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Odanacatib 50 mg OW | Placebo | Total
Number analyzed (Participants) | 8043 | 8028 | 16071
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (5.4) | 72.9 (5.3) | 72.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8043 | 8028 | 16071
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 97 | 88 | 185
  Asian | 1421 | 1411 | 2832
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 129 | 132 | 261
  White | 4528 | 4557 | 9085
  More than one race | 1867 | 1839 | 3706
  Unknown or Not Reported | 0 | 0 | 0
Stratum [Number; unit: Participants]
  Prior Vertebral Fracture | 3733 | 3737 | 7470
  No Prior Vertebral Fracture | 4310 | 4291 | 8601
Bisphosphonate-Intolerant [Number; unit: Participants]
  Yes | 1423 | 1447 | 2870
  No | 6615 | 6574 | 13189
  Data N/A | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Time From Baseline to First Morphometrically-Assessed Vertebral Fracture
Description: Morphometric vertebral fractures were assessed by central adjudication on lumbar and thoracic spinal radiographs acquired at baseline and at Months 6, 12, and subsequent yearly time points. Incident fractures (i.e., occurring after baseline) in previously normal vertebral bodies and/or those occurring after baseline in previously fractured vertebral bodies (Genant semiquantitative [SQ] Grade 1-3) (T4 to L4) were confirmed by quantitative morphometric (QM) and either SQ or binary SQ (yes/no) methodologies. A time-to-event methodology was used to evaluate results: life-table estimates of the incidence proportion (cumulative incidence) of participants with at least one morphometric vertebral fracture were assessed at Months 6, 12, and subsequent yearly intervals; an interval-censored approach was then used to determine incidence rate (number of participants with a morphometric fracture per 100 person-years of follow-up).
Time Frame: Up to approximately 60 months of observation
Population: The Full-Analysis-Set (FAS) including all randomized participants, who took at least one dose of study medication with follow-up from start of prime therapy to study termination (base study) with at least one spine radiograph on treatment (and at baseline) was used for analysis.
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6770 | 6910
Parts. w/ fracture per 100 person-years | 1.27 | 2.74
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW vs Placebo. Generalized linear model for binary data with cloglog link and terms for time interval, treatment, stratum, and geographic region. cloglog link = complementary log log transformation of probability of an event up to the time-point; Test type: Other; p < 0.001, Generalized linear model; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.40 to 0.53]

2. Primary Outcome: Base Study: Time From Baseline to First Osteoporotic Clinical Hip Fracture (Adjudicated)
Description: Osteoporotic clinical hip fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Hip fractures were fractures of the proximal femur confirmed as being located in the hip (i.e., sub-region not specified; cervical, and intertrochanteric). Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 60 months of observation
Population: The FAS including all randomized participants who took at least one dose of study medication with follow-up from start of prime therapy to study termination (base study) was used for analysis.
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. w/ fracture per 100 person-years | 0.28 | 0.54
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW vs Placebo. The Cox proportional hazards model included terms for treatment, stratum and geographic region; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.39 to 0.71]

3. Primary Outcome: Base Study: Time From Baseline to First Osteoporotic Clinical Non-Vertebral Fracture (Adjudicated)
Description: Osteoporotic non-vertebral clinical fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Non-vertebral fractures were assessed across multiple anatomical sites including clavicle, distal femur or shaft, fibula, hip, humerus, pelvis, radius, ribs, sacrum, tibia, ulna, and wrist. Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 2
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. w/ fracture per 100 person-years | 1.85 | 2.41
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.68 to 0.87]

4. Primary Outcome: Base Study + First Extension: Time From Baseline to First Morphometrically-Assessed Vertebral Fracture
Description: Morphometric vertebral fractures were confirmed by central adjudication on lumbar and thoracic spinal radiographs acquired at baseline and at Months 6, 12, and subsequent yearly time points. Incident fractures (i.e., occurring after baseline) in previously normal vertebral bodies and/or those occurring after baseline in previously fractured vertebral bodies (Genant SQ Grade 1-3) (T4 to L4) were confirmed by QM and either SQ or binary SQ (yes/no) methodologies. A time-to-event methodology was used to evaluate results: life-table estimates of the incidence proportion (cumulative incidence) of participants with at least one morphometric vertebral fracture were assessed at Months 6, 12, and subsequent yearly intervals; an interval-censored approach was then used to determine incidence rate (number of participants with a morphometric fracture per 100 person-years of follow-up).
Time Frame: Up to approximately 74 months of observation
Population: The FAS including all randomized participants, who took at least one dose of study medication with follow-up from start of prime therapy to study termination (base study + first extension-double blind period [dbp]) with at least one spine radiograph on treatment (and at baseline) was used for analysis.
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6909 | 7011
Parts. w/ fracture per 100 person-years | 1.33 | 2.74
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Generalized linear model; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.42 to 0.55]

5. Primary Outcome: Base Study + First Extension: Time From Baseline to First Osteoporotic Clinical Hip Fracture (Adjudicated)
Description: Osteoporotic clinical hip fractures was confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Hip fractures were fractures of the proximal femur confirmed as being located in the hip (i.e., sub-region not specified; cervical, and intertrochanteric). Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 74 months of observation
Population: The FAS including all randomized participants who took at least one dose of study medication with follow-up from start of prime therapy to study termination (base study + first extension-dbp) was used for analysis.
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. w/ fracture per 100 person-years | 0.29 | 0.56
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.40 to 0.67]

6. Primary Outcome: Base Study + First Extension: Time From Baseline to First Osteoporotic Clinical Non-Vertebral Fracture (Adjudicated)
Description: Osteoporotic non-vertebral clinical fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Non-vertebral fractures were assessed across multiple anatomical sites including clavicle, distal femur and shaft, fibula, hip, humerus, pelvis, radius, ribs, sacrum, tibia, ulna, and wrist. Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 5
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. w/ fracture per 100 person-years | 1.78 | 2.41
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.66 to 0.83]

7. Primary Outcome: Base Study + First Extension: Rate of Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a person or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The incidence rate of participants with adverse events (number of participants with an event per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 74 months of observation
Population: The All-Participants-as-Treated population including all randomized participants who took at least one dose of study medication was used for analysis (base study + first extension).
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 97.25 [95.00 to 99.53] | 96.36 [94.13 to 98.63]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.88, 95% CI 2-sided [-2.3 to 4.07]

8. Primary Outcome: Base Study + First Extension: Rate of Discontinuations From Study Treatment Due to an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a person or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The incidence rate of participant discontinuations from treatment due to adverse events (number of participants with an event per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 2.66 [2.48 to 2.86] | 2.55 [2.37 to 2.75]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.11, 95% CI 2-sided [-0.16 to 0.37]

9. Primary Outcome: Base Study + First Extension + Second Extension: Percent Change From Baseline in Bone Mineral Density (BMD) Measurements of the Total Hip
Description: BMD was measured by dual-energy x-ray absorptiometry (DXA) at the total hip starting at screening, and at yearly intervals until the end of the study (second extension study) for all participants who entered the second extension study. Least squares (LS) means percent change in BMD from original baseline are provided through Month 108 (Year 9). At Months 96 (Year 8) and 108 (Year 9), approximately 3% or fewer participants in each treatment group had BMD data, and results at those time points should be viewed with caution. NOTE: The mean percent change in BMD from baseline in participants originally randomized to placebo includes BMD results obtained after those participants were switched to open-label odanacatib, which occurred at different times relative to their start of blinded study medication in the base study.
Time Frame: Baseline and once yearly, up to approximately 108 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (total hip BMD) was used for analysis (base study + first extension-dbp + second extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo: Participants received blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 2997 | 2212
Percent change
  Month 12 | 3.03 [2.91 to 3.14] | 1.08 [0.95 to 1.22]
  Month 24: number analyzed (Participants) | 2965 | 2189
  Month 24 | 4.32 [4.18 to 4.46] | 0.58 [0.42 to 0.74]
  Month 36: number analyzed (Participants) | 2950 | 2171
  Month 36 | 5.60 [5.43 to 5.77] | 0.04 [-0.16 to 0.24]
  Month 48: number analyzed (Participants) | 2905 | 2133
  Month 48 | 6.56 [6.36 to 6.76] | -0.74 [-0.97 to -0.51]
  Month 60: number analyzed (Participants) | 2718 | 2015
  Month 60 | 7.45 [7.22 to 7.68] | -1.40 [-1.67 to -1.13]
  Month 72: number analyzed (Participants) | 2186 | 1637
  Month 72 | 7.88 [7.62 to 8.14] | -0.01 [-0.31 to 0.30]
  Month 84: number analyzed (Participants) | 1631 | 1197
  Month 84 | 7.94 [7.63 to 8.26] | 0.97 [0.61 to 1.34]
  Month 96: number analyzed (Participants) | 237 | 187
  Month 96 | 7.87 [7.38 to 8.37] | 1.57 [1.01 to 2.13]
  Month 108: number analyzed (Participants) | 63 | 51
  Month 108 | 7.03 [6.02 to 8.05] | 1.11 [-0.02 to 2.23]

10. Primary Outcome: Second Extension: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a person or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to approximately 34 months of observation
Population: The All-Participants-as-Treated population including all randomized participants who took at least one dose of study medication was used for the analysis (second extension study).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Originally Assigned to Placebo): Participants received blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for up to 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Arm/Group | Odanacatib 50 mg OW | Placebo (Originally Assigned to Placebo)
Number analyzed (Participants) | 3144 | 2309
Participants | 2173 | 1587

11. Primary Outcome: Second Extension: Number of Participants Discontinuing Study Treatment Due to an Adverse Event
Description: as for outcome 10
Time Frame: Up to approximately 34 months of observation
Population: The All-Participants-as-Treated population including all randomized participants who took at least one dose of study medication was used for analysis (second extension study).
Measure: Count of Participants; unit: Participants
Arm/Group | Odanacatib 50 mg OW | Placebo (Originally Assigned to Placebo)
Number analyzed (Participants) | 3144 | 2309
Participants | 55 | 36

12. Primary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in Volumetric Bone Mineral Density (vBMD) at the Lumbar Spine Using Quantitative Computed Tomography
Description: Compartment-specific effects of osteoporosis were assessed by measuring trabecular vBMD at the lumbar spine (L1 total vertebral body) using quantitative computed tomography. The percent change from baseline at Month 24 (base study) was then assessed using a longitudinal data analysis model including terms for treatment, stratum (prior vertebral fracture [yes/no]) and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (lumbar spine vBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 46 | 48
Percent change | 8.05 [4.48 to 11.62] | -0.87 [-4.37 to 2.64]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg vs Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.92, 95% CI 2-sided [3.9 to 13.93]

13. Primary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in vBMD at the Lumbar Spine Using Quantitative Computed Tomography
Description: Compartment-specific effects of osteoporosis were assessed by measuring trabecular vBMD at the lumbar spine (L1 total vertebral body) using quantitative computed tomography. The percent change from baseline at Month 60 (base study + extension study) was then assessed using a longitudinal data analysis model including terms for treatment, stratum (prior vertebral fracture [yes/no]) and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (lumbar spine vBMD) was used for analysis (PN032-Base + Extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 28 | 25
Percent change | 14.76 [7.68 to 21.83] | -11.69 [-18.69 to -4.69]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg vs Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 26.45, 95% CI 2-sided [16.49 to 36.40]

14. Primary Outcome: Sarcopenia Substudy PN035: Change From Baseline in Appendicular Lean Body Mass (aLBM)
Description: Sarcopenia is the age-related loss of skeletal muscle mass and associated loss of strength. Progression of sarcopenia was assessed using aLBM as measured by total body DXA. The change from baseline at yearly intervals was then assessed using a longitudinal data analysis model with terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline and once yearly up to 4 years
Population: The FAS for change from baseline at specific time-points including all randomized participants who took at least one dose of study medication and had the necessary baseline and on-treatment measurements available (aLBM) was used for analysis (PN035).
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 247 | 257
kg
  Month 12 | -0.20 [-0.28 to -0.12] | -0.18 [-0.26 to -0.10]
  Month 24: number analyzed (Participants) | 239 | 236
  Month 24 | -0.19 [-0.28 to -0.10] | -0.19 [-0.28 to -0.10]
  Month 36: number analyzed (Participants) | 201 | 187
  Month 36 | -0.36 [-0.45 to -0.27] | -0.32 [-0.41 to -0.23]
  Month 48: number analyzed (Participants) | 36 | 32
  Month 48 | -0.44 [-0.64 to -0.24] | -0.23 [-0.44 to -0.02]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12. Longitudinal model includes terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size); Test type: Other; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.14 to 0.09]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24. Longitudinal model includes terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size); Test type: Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.12 to 0.12]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36. Longitudinal model includes terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size); Test type: Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.17 to 0.09]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48. Longitudinal model includes terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size); Test type: Other; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.50 to 0.08]

15. Primary Outcome: Sarcopenia Substudy PN035: Change From Baseline in Short Physical Performance Battery (SPPB) Score
Description: The Short Physical Performance Battery (SPPB) Score is used to assess physical function in older persons. The SPPB consists of 3 types of physical activities: standing balance, gait speed, and chair rise. Component activities are timed and then reduced to a categorical 0 to 4 scale based on time achieved. A higher composite score (range 0 to 12) indicates an improved function level. The change from baseline at yearly intervals was then assessed using a longitudinal data analysis model with terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline and once yearly up to 4 years
Population: The FAS for change from baseline at specific time-points including all randomized participants who took at least one dose of study medication and had the necessary baseline and on-treatment measurements available (SPPB) was used for analysis (PN035).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 251 | 253
Score on a scale
  Month 12 | 0.03 [-0.16 to 0.22] | -0.08 [-0.27 to 0.11]
  Month 24: number analyzed (Participants) | 248 | 235
  Month 24 | -0.04 [-0.25 to 0.16] | -0.19 [-0.40 to 0.02]
  Month 36: number analyzed (Participants) | 230 | 221
  Month 36 | -0.18 [-0.42 to 0.06] | -0.37 [-0.62 to -0.13]
  Month 48: number analyzed (Participants) | 136 | 111
  Month 48 | -0.05 [-0.34 to 0.24] | -0.24 [-0.55 to 0.07]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Other; Difference in Least Squares Means = 0.11, 95% CI 2-sided [-0.16 to 0.38]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Other; Difference in Least Squares Means = 0.14, 95% CI 2-sided [-0.15 to 0.44]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Other; Difference in Least Squares Means = 0.19, 95% CI 2-sided [-0.15 to 0.54]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Other; Difference in Least Squares Means = 0.19, 95% CI 2-sided [-0.24 to 0.62]

16. Primary Outcome: Sarcopenia Substudy PN035: Change From Baseline in Gait Speed
Description: Gait speed is a component of the Short Physical Performance Battery (SPPB) Score. Participants are asked to walk a distance of 4 meters at their normal pace. The test is performed 2 times, and the walk done in the shortest time is used for scoring. The activity is timed and then reduced to a categorical 0 to 4 scale based on time achieved. Higher scores indicate an improved function level. The change from baseline at yearly intervals was then assessed using a longitudinal data analysis model with terms for treatment, stratum (sarcopenia, non-sarcopenia), time and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline and once yearly up to 4 years.
Population: The FAS for change from baseline at specific time-points including all randomized participants who took at least one dose of study medication and had the necessary baseline and on-treatment measurements available (gait speed) was used for analysis (PN035).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Placebo: Participants receive blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for up to 5 years. Participants also receive Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) is approximately 1200 mg.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 249 | 252
Score on a scale
  Month 12 | -0.02 [-0.10 to 0.06] | -0.06 [-0.14 to 0.02]
  Month 24: number analyzed (Participants) | 245 | 233
  Month 24 | -0.02 [-0.11 to 0.07] | -0.10 [-0.19 to -0.00]
  Month 36: number analyzed (Participants) | 227 | 218
  Month 36 | -0.09 [-0.19 to 0.02] | -0.11 [-0.22 to -0.01]
  Month 48: number analyzed (Participants) | 135 | 111
  Month 48 | -0.15 [-0.28 to -0.02] | -0.24 [-0.38 to -0.10]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Other; Difference in Least Squares Means = 0.04, 95% CI 2-sided [-0.08 to 0.15]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Other; Difference in Least Squares Means = 0.08, 95% CI 2-sided [-0.06 to 0.21]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Other; Difference in Least Squares Means = 0.03, 95% CI 2-sided [-0.12 to 0.17]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Other; Difference in Least Squares Means = 0.09, 95% CI 2-sided [-0.09 to 0.28]

17. Secondary Outcome: Base Study: Rate of Adverse Events
Description: as for outcome 7
Time Frame: Up to approximately 60 months of observation
Population: The All-Participants-as-Treated population including all randomized participants who took at least one dose of study medication was used for analysis (base study).
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 100.16 [97.81 to 102.6] | 98.65 [96.33 to 101.01]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 1.52, 95% CI 2-sided [-1.8 to 4.84]

18. Secondary Outcome: Base Study: Rate of Discontinuation From Study Treatment Due to an Adverse Event
Description: as for outcome 8
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 2.97 [2.75 to 3.20] | 2.70 [2.49 to 2.92]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.27, 95% CI 2-sided [-0.04 to 0.58]

19. Secondary Outcome: Base Study: Time From Baseline to First Osteoporotic Clinical Vertebral Fracture (Adjudicated)
Description: Osteoporotic vertebral clinical fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Vertebral fractures were assessed for all vertebral levels (C7, T1 to T12, L1 to L5). Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 2
Measure: Number; unit: Parts. w/ fracture per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. w/ fracture per 100 person-years | 0.16 | 0.58
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.19 to 0.40]

20. Secondary Outcome: Base Study: Yearly Rate of Height Loss
Description: Height was measured by wall-mounted stadiometer at randomization and at yearly intervals in the base study.
Time Frame: Up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (height) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6112 | 6231
cm/year | -0.13 [-0.14 to -0.12] | -0.15 [-0.16 to -0.14]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW versus Placebo. The mixed model contained fixed effects for treatment, region, stratum, treatment-year interaction and random effect intercept and slope (year) and unstructured covariance matrix; Test type: Other; p = 0.041, Mixed Models Analysis; Difference in Least Squares Means = 0.01, 95% CI 2-sided [0.00 to 0.03]

21. Secondary Outcome: Base Study: Number of Participants With Height Loss of > 1 cm
Description: Height was measured by wall-mounted stadiometer at randomization and at yearly intervals in the base study.
Time Frame: Baseline and once yearly, up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (height loss) was used for analysis (base study).
Measure: Count of Participants; unit: Participants
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6095 | 6215
Participants
  Up to Month 12 | 316 | 365
  Up to Month 24: number analyzed (Participants) | 5347 | 5396
  Up to Month 24 | 592 | 669
  Up to Month 36: number analyzed (Participants) | 4745 | 4632
  Up to Month 36 | 875 | 944
  Up to Month 48: number analyzed (Participants) | 331 | 281
  Up to Month 48 | 90 | 59
  Up to Month 60: number analyzed (Participants) | 103 | 70
  Up to Month 60 | 23 | 12
  Overall/At any time | 1022 | 1149
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW versus Placebo. Treatment comparison for height loss at any time during the treatment period. The logistic model contained terms for treatment, geographic region and stratum; Test type: Other; p = 0.014, Logistic model; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.81 to 0.98]

22. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Total Hip
Description: BMD was measured by DXA for all participants at the total hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (total hip BMD) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6490 | 6596
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 1.85 [1.54 to 2.16] | 0.53 [0.24 to 0.81]
  Month 12 | 2.82 [2.74 to 2.91] | 0.33 [0.25 to 0.42]
  Month 24: number analyzed (Participants) | 5916 | 5895
  Month 24 | 3.79 [3.68 to 3.90] | -0.68 [-0.79 to -0.57]
  Month 36: number analyzed (Participants) | 5127 | 4925
  Month 36 | 4.81 [4.67 to 4.94] | -1.64 [-1.78 to -1.50]
  Month 48: number analyzed (Participants) | 539 | 452
  Month 48 | 5.39 [5.04 to 5.74] | -3.23 [-3.59 to -2.87]
  Month 60: number analyzed (Participants) | 167 | 138
  Month 60 | 5.67 [5.13 to 6.21] | -3.82 [-4.40 to -3.24]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 6. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.32, 95% CI 2-sided [0.90 to 1.75]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.49, 95% CI 2-sided [2.37 to 2.61]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.47, 95% CI 2-sided [4.31 to 4.62]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.44, 95% CI 2-sided [6.25 to 6.64]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.62, 95% CI 2-sided [8.11 to 9.12]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 60. The longitudinal model includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.49, 95% CI 2-sided [8.70 to 10.29]

23. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Lumbar Spine
Description: BMD was measured by DXA for all participants at the lumbar spine at randomization, Months 6, 12, and subsequent yearly intervals until the end of the study (base study). Measurements were made on at least 3 vertebrae for all time points; vertebrae with fractures were excluded from analyses.
  at
Time Frame: Baseline, Month 6, and once yearly, approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (lumbar spine BMD) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6344 | 6400
Percent change
  Month 6: number analyzed (Participants) | 293 | 299
  Month 6 | 3.75 [3.39 to 4.11] | 0.78 [0.44 to 1.13]
  Month 12 | 4.67 [4.56 to 4.77] | 0.59 [0.49 to 0.70]
  Month 24: number analyzed (Participants) | 5805 | 5778
  Month 24 | 6.77 [6.64 to 6.90] | 0.72 [0.59 to 0.84]
  Month 36: number analyzed (Participants) | 5086 | 4913
  Month 36 | 8.59 [8.43 to 8.74] | 0.75 [0.59 to 0.90]
  Month 48: number analyzed (Participants) | 503 | 441
  Month 48 | 10.47 [10.09 to 10.86] | 0.76 [0.35 to 1.16]
  Month 60: number analyzed (Participants) | 169 | 138
  Month 60 | 11.49 [10.82 to 12.17] | 0.26 [-0.47 to 1.00]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.96, 95% CI 2-sided [2.47 to 3.46]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.07, 95% CI 2-sided [3.93 to 4.22]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.05, 95% CI 2-sided [5.87 to 6.23]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 7.84, 95% CI 2-sided [7.62 to 8.06]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.72, 95% CI 2-sided [9.16 to 10.27]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 11.23, 95% CI 2-sided [10.23 to 12.23]

24. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Femoral Neck
Description: BMD was measured by DXA for all participants at the femoral neck-hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (femoral neck BMD) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6490 | 6597
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 2.17 [1.78 to 2.55] | 0.68 [0.30 to 1.06]
  Month 12 | 2.80 [2.68 to 2.91] | 0.59 [0.48 to 0.70]
  Month 24: number analyzed (Participants) | 5916 | 5895
  Month 24 | 4.01 [3.88 to 4.15] | -0.37 [-0.50 to -0.23]
  Month 36: number analyzed (Participants) | 5126 | 4925
  Month 36 | 5.45 [5.29 to 5.61] | -1.01 [-1.17 to -0.85]
  Month 48: number analyzed (Participants) | 539 | 452
  Month 48 | 6.15 [5.74 to 6.56] | -2.27 [-2.71 to -1.83]
  Month 60: number analyzed (Participants) | 167 | 138
  Month 60 | 6.69 [6.02 to 7.36] | -1.84 [-2.58 to -1.11]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.49, 95% CI 2-sided [0.95 to 2.03]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.21, 95% CI 2-sided [2.05 to 2.37]
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.38, 95% CI 2-sided [4.19 to 4.57]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.46, 95% CI 2-sided [6.24 to 6.68]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.42, 95% CI 2-sided [7.82 to 9.02]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.53, 95% CI 2-sided [7.54 to 9.53]

25. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Trochanter
Description: BMD was measured by DXA for all participants at the trochanter-hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (trochanter BMD) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6490 | 6596
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 2.65 [2.12 to 3.18] | 0.91 [0.43 to 1.38]
  Month 12 | 4.32 [4.18 to 4.46] | 0.82 [0.68 to 0.96]
  Month 24: number analyzed (Participants) | 5916 | 5895
  Month 24 | 6.17 [6.00 to 6.34] | -0.24 [-0.41 to -0.07]
  Month 36: number analyzed (Participants) | 5127 | 4925
  Month 36 | 8.01 [7.81 to 8.22] | -1.26 [-1.47 to -1.05]
  Month 48: number analyzed (Participants) | 539 | 452
  Month 48 | 9.46 [8.92 to 10.00] | -2.98 [-3.54 to -2.42]
  Month 60: number analyzed (Participants) | 167 | 138
  Month 60 | 10.16 [9.32 to 10.99] | -3.65 [-4.55 to -2.75]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.74, 95% CI 2-sided [1.03 to 2.46]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 3.50, 95% CI 2-sided [3.31 to 3.70]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24; Test type: Other; p < 0.001, Longitudinal model; Includes terms for treatment, stratum, region & interaction between treatment & time as fixed effects (LS means weighted for region & stratum size); Difference in Least Squares Means = 6.41, 95% CI 2-sided [6.17 to 6.65]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 9.27, 95% CI 2-sided [8.98 to 9.57]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 12.44, 95% CI 2-sided [11.66 to 13.22]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 60; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 13.81, 95% CI 2-sided [12.58 to 15.04]

26. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Distal-Third Forearm
Description: BMD was measured by DXA at the distal one-third radius at randomization and at yearly intervals until the end of the study (base study) in an approximate 10% random subset of participants at selected sites.
Time Frame: Baseline and once yearly, up to approximately 60 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (distal one-third radius BMD) was used for analysis (base study).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 679 | 718
Percent change
  Month 12 | 0.51 [0.19 to 0.82] | -0.60 [-0.91 to -0.30]
  Month 24: number analyzed (Participants) | 615 | 635
  Month 24 | 0.33 [-0.03 to 0.68] | -1.02 [-1.37 to -0.68]
  Month 36: number analyzed (Participants) | 569 | 558
  Month 36 | 0.02 [-0.36 to 0.41] | -1.90 [-2.29 to -1.52]
  Month 48: number analyzed (Participants) | 85 | 77
  Month 48 | -0.62 [-1.52 to 0.28] | -2.82 [-3.76 to -1.88]
  Month 60: number analyzed (Participants) | 32 | 26
  Month 60 | 0.29 [-1.08 to 1.66] | -3.21 [-4.72 to -1.70]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.11, 95% CI 2-sided [0.67 to 1.55]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.35, 95% CI 2-sided [0.85 to 1.84]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.93, 95% CI 2-sided [1.38 to 2.47]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p = 0.001, Longitudinal model; Difference in Least Squares Means = 2.20, 95% CI 2-sided [0.89 to 3.51]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p = 0.001, Longitudinal model; Difference in Least Squares Means = 3.50, 95% CI 2-sided [1.46 to 5.54]

27. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Lumbar Spine in Bisphosphonate-Intolerant Participants
Description: BMD was measured by DXA in bisphosphonate-intolerant participants at the lumbar spine at randomization, and at yearly intervals until the end of the study (base study). Measurements were made on at least 3 vertebrae for all time points; vertebrae with fractures were excluded from analyses. Bisphosphonates are anti-resorptive agents used in the treatment of osteoporosis. Bisphosphonate-intolerance was defined by contraindication or history of intolerance to bisphosphonates, or physician's determination of unsuitability for bisphosphonate treatment.
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: as for outcome 23
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 1116 | 1127
Percent change
  Month 6: number analyzed (Participants) | 26 | 32
  Month 6 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
  Month 12 | 4.56 [4.31 to 4.80] | 0.54 [0.29 to 0.78]
  Month 24: number analyzed (Participants) | 1025 | 1004
  Month 24 | 6.60 [6.31 to 6.90] | 0.82 [0.52 to 1.11]
  Month 36: number analyzed (Participants) | 889 | 853
  Month 36 | 8.49 [8.13 to 8.85] | 0.87 [0.50 to 1.23]
  Month 48: number analyzed (Participants) | 63 | 40
  Month 48 | 10.31 [9.34 to 11.29] | 0.80 [-0.40 to 2.00]
  Month 60: number analyzed (Participants) | 2 | 9
  Month 60 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 5.79, 95% CI 2-sided [5.37 to 6.2]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.02, 95% CI 2-sided [3.67 to 4.37]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 7.62, 95% CI 2-sided [7.11 to 8.13]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.51, 95% CI 2-sided [7.96 to 11.06]

28. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Total Hip in Bisphosphonate-Intolerant Participants
Description: BMD was measured by DXA in bisphosphonate-intolerant participants at the total hip at screening, and at yearly intervals until the end of the study (base study). Bisphosphonates are anti-resorptive agents used in the treatment of osteoporosis. Bisphosphonate-intolerance was defined by contraindication or history of intolerance to bisphosphonates, or physician's determination of unsuitability for bisphosphonate treatment.
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: as for outcome 22
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 1127 | 1155
Percent change
  Month 6: number analyzed (Participants) | 25 | 34
  Month 6 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
  Month 12 | 2.63 [2.43 to 2.83] | 0.24 [0.04 to 0.44]
  Month 24: number analyzed (Participants) | 1035 | 1020
  Month 24 | 3.56 [3.30 to 3.82] | -0.64 [-0.90 to -0.39]
  Month 36: number analyzed (Participants) | 889 | 853
  Month 36 | 4.45 [4.14 to 4.76] | -1.41 [-1.72 to -1.09]
  Month 48: number analyzed (Participants) | 65 | 42
  Month 48 | 4.07 [3.09 to 5.04] | -4.47 [-5.67 to -3.27]
  Month 60: number analyzed (Participants) | 2 | 10
  Month 60 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.40, 95% CI 2-sided [2.11 to 2.68]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.21, 95% CI 2-sided [3.84 to 4.57]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 5.86, 95% CI 2-sided [5.41 to 6.30]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.54, 95% CI 2-sided [7.00 to 10.09]

29. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Femoral Neck in Bisphosphonate-Intolerant Participants
Description: BMD was measured by DXA in bisphosphonate-intolerant participants at the femoral neck-hip at screening, and at yearly intervals until the end of the study (base study). Bisphosphonates are anti-resorptive agents used in the treatment of osteoporosis. Bisphosphonate-intolerance was defined by contraindication or history of intolerance to bisphosphonates, or physician's determination of unsuitability for bisphosphonate treatment.
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 1127 | 1156
Percent change
  Month 6: number analyzed (Participants) | 25 | 34
  Month 6 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
  Month 12 | 2.71 [2.44 to 2.98] | 0.50 [0.24 to 0.77]
  Month 24: number analyzed (Participants) | 1035 | 1020
  Month 24 | 3.88 [3.56 to 4.19] | -0.45 [-0.77 to -0.13]
  Month 36: number analyzed (Participants) | 889 | 853
  Month 36 | 5.12 [4.75 to 5.50] | -0.97 [-1.35 to -0.59]
  Month 48: number analyzed (Participants) | 65 | 42
  Month 48 | 6.75 [5.43 to 8.08] | -2.32 [-3.96 to -0.68]
  Month 60: number analyzed (Participants) | 2 | 10
  Month 60 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.21, 95% CI 2-sided [1.83 to 2.59]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.33, 95% CI 2-sided [3.87 to 4.78]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.09, 95% CI 2-sided [5.56 to 6.62]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.08, 95% CI 2-sided [6.97 to 11.19]

30. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Trochanter in Bisphosphonate-Intolerant Participants
Description: BMD was measured by DXA in bisphosphonate-intolerant participants at the trochanter-hip at screening, and at yearly intervals until the end of the study (base study). Bisphosphonates are anti-resorptive agents used in the treatment of osteoporosis. Bisphosphonate-intolerance was defined by contraindication or history of intolerance to bisphosphonates, or physician's determination of unsuitability for bisphosphonate treatment.
Time Frame: Baseline, Month 6, and once yearly, up to approximately 60 months of observation
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 1127 | 1155
Percent change
  Month 6: number analyzed (Participants) | 25 | 34
  Month 6 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
  Month 12 | 4.02 [3.70 to 4.35] | 0.58 [0.26 to 0.90]
  Month 24: number analyzed (Participants) | 1035 | 1020
  Month 24 | 5.73 [5.33 to 6.12] | -0.30 [-0.70 to 0.10]
  Month 36: number analyzed (Participants) | 889 | 853
  Month 36 | 7.47 [6.99 to 7.94] | -1.02 [-1.50 to -0.54]
  Month 48: number analyzed (Participants) | 65 | 42
  Month 48 | 6.68 [5.04 to 8.32] | -5.07 [-7.09 to -3.05]
  Month 60: number analyzed (Participants) | 2 | 10
  Month 60 | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model. | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 3.44, 95% CI 2-sided [2.98 to 3.90]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.03, 95% CI 2-sided [5.47 to 6.59]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.49, 95% CI 2-sided [7.81 to 9.16]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 11.76, 95% CI 2-sided [9.15 to 14.36]

31. Secondary Outcome: Base Study: Percent Change From Baseline in BMD Measurements of the Distal-Third Forearm in Bisphosphonate-Intolerant Participants
Description: BMD was measured by DXA at the distal one-third radius at randomization and at yearly intervals until the end of the study (base study) in an approximate 10% random subset of bisphosphonate-intolerant participants at selected sites. Bisphosphonates are anti-resorptive agents used in the treatment of osteoporosis. Bisphosphonate-intolerance was defined by contraindication or history of intolerance to bisphosphonates, or physician's determination of unsuitability for bisphosphonate treatment.
Time Frame: Baseline and once yearly, up to approximately 60 months of observation
Population: as for outcome 26
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 77 | 112
Percent change
  Month 12 | 0.99 [0.06 to 1.93] | -0.09 [-0.87 to 0.69]
  Month 24: number analyzed (Participants) | 71 | 100
  Month 24 | 0.24 [-0.79 to 1.28] | -0.80 [-1.67 to 0.06]
  Month 36: number analyzed (Participants) | 64 | 82
  Month 36 | -0.66 [-1.76 to 0.44] | -1.87 [-2.82 to -0.92]
  Month 48: number analyzed (Participants) | 8 | 5
  Month 48 | -0.72 [-4.90 to 3.45] | -2.27 [-7.23 to 2.68]
  Month 60: number analyzed (Participants) | 0 | 2
  Month 60 |  | NA [NA to NA] — Not calculated due to convergence issue with longitudinal data analysis model.
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p = 0.083, Longitudinal model; Difference in Least Squares Means = 1.08, 95% CI 2-sided [-0.14 to 2.31]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p = 0.129, Longitudinal model; Difference in Least Squares Means = 1.05, 95% CI 2-sided [-0.31 to 2.40]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p = 0.104, Longitudinal model; Difference in Least Squares Means = 1.21, 95% CI 2-sided [-0.25 to 2.67]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p = 0.617, Longitudinal model; Difference in Least Squares Means = 1.55, 95% CI 2-sided [-4.92 to 8.02]

32. Secondary Outcome: Base Study: Percent Change From Baseline in Serum C-Telopeptides of Type I Collagen (s-CTx) After Log-Transformation
Description: s-CTx, a biochemical marker of bone resorption by osteoclasts reflecting collagen breakdown products, was assessed at randomization, Month 6, and at yearly intervals until the end of the study (base study) in an approximate 10% random subset participants at selected sites. The log-transformed fraction from baseline in s-CTx was determined using a longitudinal model with terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS means weighted for region and stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 6, and once yearly up to 4 years
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (s-CTx) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (base study).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 618 | 629
Percent change
  Month 6: number analyzed (Participants) | 571 | 585
  Month 6 | -61.27 [-63.33 to -59.09] | -2.28 [-7.43 to 3.15]
  Month 12 | -53.47 [-55.98 to -50.81] | 6.54 [0.85 to 12.56]
  Month 24: number analyzed (Participants) | 528 | 534
  Month 24 | -39.47 [-42.61 to -36.15] | 7.23 [1.70 to 13.07]
  Month 36: number analyzed (Participants) | 447 | 414
  Month 36 | -23.71 [-27.79 to -19.40] | 20.96 [14.38 to 27.91]
  Month 48: number analyzed (Participants) | 528 | 534
  Month 48 | -4.61 [-15.93 to 8.24] | 14.12 [0.47 to 29.61]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 6; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -58.99, 95% CI 2-sided [-64.68 to -53.30]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -60.01, 95% CI 2-sided [-66.40 to -53.61]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -46.70, 95% CI 2-sided [-53.23 to -40.17]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36; Test type: Other; p = 0.050, Longitudinal model; Difference in Least Squares Means = -44.67, 95% CI 2-sided [-52.62 to -36.72]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48; Test type: Other; p = 0.050, Longitudinal model; Difference in Least Squares Means = -18.73, 95% CI 2-sided [-37.44 to -0.01]

33. Secondary Outcome: Base Study: Percent Change From Baseline in Urinary N-Telopeptides of Type I Collagen/Creatinine (u-NTx/Cr) Ratio After Log-Transformation
Description: u-NTx, a biochemical marker of bone resorption, was assessed at randomization, Month 6, and at yearly intervals until the end of the study (base study) in an approximate 10% random subset participants at selected sites. Urine NTx measurements (in bone collagen equivalents [BCE]) were normalized to urine Cr concentration (i.e., u-NTx/Cr ratio) and the log-transformed fraction from baseline in u-NTx/Cr ratio was then determined using a longitudinal model with terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS means weighted for region and stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 6, and once yearly up to 4 years
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (u-NTx/Cr) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (base study).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Groups:
- Odanacatib 50 mg OW: Participants received 50 mg of blinded odanacatib weekly over the course of the base study and first extension study (5 years total), followed by 50 mg of open-label odanacatib weekly for 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
- Placebo: Participants received blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total), followed by 50 mg of open-label odanacatib weekly for 5 years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 603 | 619
Percent change
  Month 6: number analyzed (Participants) | 554 | 569
  Month 6 | -56.46 [-58.27 to -54.56] | -4.76 [-8.68 to -0.67]
  Month 12 | -55.58 [-57.54 to -53.53] | -1.99 [-6.26 to 2.48]
  Month 24: number analyzed (Participants) | 516 | 516
  Month 24 | -47.21 [-49.70 to -44.61] | 9.46 [4.33 to 14.85]
  Month 36: number analyzed (Participants) | 438 | 406
  Month 36 | -43.91 [-46.80 to -40.86] | 15.23 [9.15 to 21.64]
  Month 48: number analyzed (Participants) | 49 | 52
  Month 48 | -38.01 [-46.30 to -28.43] | 6.53 [-7.38 to 22.53]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 6; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -51.70, 95% CI 2-sided [-56.11 to -47.28]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -53.59, 95% CI 2-sided [-58.39 to -48.79]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -56.68, 95% CI 2-sided [-62.52 to -50.84]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -59.14, 95% CI 2-sided [-66.04 to -52.23]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -44.54, 95% CI 2-sided [-61.72 to -27.36]

34. Secondary Outcome: Base Study: Percent Change From Baseline in Bone-Specific Alkaline Phosphatase (BSAP) After Log-Transformation
Description: BSAP is an enzyme produced by matrix-synthesizing osteoblasts during the synthesis of collagenous bone matrix (type 1 collagen) used as a biochemical marker of bone formation. Serum BSAP was assessed at randomization, Month 6, and at yearly intervals until the end of the study (base study) in an approximate 10% random subset participants at selected sites. The log-transformed fraction from baseline in BSAP was determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 6, and once yearly up to 4 years
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (BSAP) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (base study).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 634 | 650
Percent change
  Month 6: number analyzed (Participants) | 594 | 614
  Month 6 | -23.27 [-25.12 to -21.38] | -9.13 [-11.28 to -6.93]
  Month 12 | -21.43 [-23.53 to -19.27] | -9.42 [-11.80 to -6.97]
  Month 24: number analyzed (Participants) | 543 | 545
  Month 24 | -9.33 [-12.10 to -6.47] | -0.04 [-3.07 to 3.08]
  Month 36: number analyzed (Participants) | 460 | 433
  Month 36 | -8.41 [-11.23 to -5.51] | -0.77 [-3.85 to 2.40]
  Month 48: number analyzed (Participants) | 59 | 55
  Month 48 | -0.63 [-8.39 to 7.80] | 0.15 [-7.93 to 8.94]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 6. Longitudinal model includes terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS Means weighted for region and stratum size); Test type: Other; p < 0.001, Longitudinal model; Mean Difference (Final Values) = -14.13, 95% CI 2-sided [-17.00 to -11.27]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 12. Longitudinal model includes terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS Means weighted for region and stratum size); Test type: Other; p < 0.001, Longitudinal model; Mean Difference (Final Values) = -12.01, 95% CI 2-sided [-15.22 to -8.79]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24. Longitudinal model includes terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS Means weighted for region and stratum size); Test type: Other; p < 0.001, Longitudinal model; Mean Difference (Final Values) = -9.29, 95% CI 2-sided [-13.45 to -5.13]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 36. Longitudinal model includes terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS Means weighted for region and stratum size); Test type: Other; p < 0.001, Longitudinal model; Mean Difference (Final Values) = -7.64, 95% CI 2-sided [-11.87 to -3.41]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 48. Longitudinal model includes terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS Means weighted for region and stratum size); Test type: Other; p = 0.896, Longitudinal model; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-12.34 to 10.79]

35. Secondary Outcome: Base Study: Percent Change From Baseline in N-Terminal Propeptide of Type 1 Collagen (P1NP) After Log-Transformation
Description: P1NP is a cleavage fragment produced during the synthesis of collagenous bone matrix (type 1 collagen) used as a biochemical marker of bone formation. Serum P1NP was assessed at randomization, Month 6, and at yearly intervals until the end of the study (base study) in an approximate 10% random subset participants at selected sites. The log-transformed fraction from baseline in P1NP was determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 6, and once yearly up to 4 years
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (P1NP) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (base study).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 634 | 650
Percent change
  Month 6: number analyzed (Participants) | 594 | 613
  Month 6 | -44.51 [-46.71 to -42.23] | -15.08 [-18.39 to -11.65]
  Month 12 | -37.49 [-40.12 to -34.75] | -11.55 [-15.21 to -7.72]
  Month 24: number analyzed (Participants) | 534 | 545
  Month 24 | -22.46 [-25.69 to -19.09] | -6.20 [-10.08 to -2.16]
  Month 36: number analyzed (Participants) | 460 | 433
  Month 36 | -11.89 [-15.70 to -7.92] | 0.22 [-4.15 to 4.78]
  Month 48: number analyzed (Participants) | 59 | 55
  Month 48 | -3.61 [-12.04 to 5.62] | -0.28 [-9.25 to 9.58]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 34, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Mean Difference (Final Values) = -29.43, 95% CI 2-sided [-33.47 to -25.39]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 34, analysis 2]; Test type: Other; p < 0.001, Longitudinal; Mean Difference (Final Values) = -25.94, 95% CI 2-sided [-30.54 to -21.34]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 34, analysis 3]; Test type: Other; p < 0.001, Longitudinal; Mean Difference (Final Values) = -16.26, 95% CI 2-sided [-21.41 to -11.12]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 34, analysis 4]; Test type: Other; p < 0.001, Longitudinal; Mean Difference (Final Values) = -12.11, 95% CI 2-sided [-18.03 to -6.19]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 34, analysis 5]; Test type: Other; p = 0.610, Longitudinal; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-16.12 to 9.45]

36. Secondary Outcome: Base Study: Time to First 3-Point Major Adverse Cardiac Event (MACE) Confirmed by Thrombolysis in Myocardial Infarction Study Group (TIMI) Adjudication
Description: The time to first TIMI-adjudicated 3-point MACE (a composite outcome measure of 1. cardiovascular death, 2. non-fatal definite MI, or 3. non-fatal definite stroke) was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.17 | 1.04
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.182, Regression, Cox; No adjustments for multiplicity were applied; p-value is unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.95 to 1.34]

37. Secondary Outcome: Base Study: Time to First New Onset Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated new or presumed new onset atrial fibrillation or atrial flutter was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Participants with known history of atrial fibrillation or atrial flutter were excluded and electrocardiogram confirmation was not required. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.48 | 0.41
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.235, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.9 to 1.55]

38. Secondary Outcome: Base Study: Time to First 4-Point MACE Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated 4-point MACE (a composite outcome measure of 1. cardiovascular death, 2. non-fatal definite MI, 3. non-fatal definite stroke, or 4. hospitalization for unstable angina) was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.28 | 1.14
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.127, Regression, Cox; No adjustments for multiplicity were applied; p-value is unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.97 to 1.29]

39. Secondary Outcome: Base Study: Time to First Hospitalization for Unstable Angina Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated hospitalization for unstable angina was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.10 | 0.09
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.857, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.59 to 1.89]

40. Secondary Outcome: Base Study: Time to First New Onset ECG-Confirmed Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated new or presumed new onset atrial fibrillation or atrial flutter was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Participants with known history of atrial fibrillation or atrial flutter were excluded and electrocardiogram confirmation was required. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.25 | 0.23
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.606, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.76 to 1.59]

41. Secondary Outcome: Base Study: Time to First Any Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated any reported episode of atrial fibrillation or atrial flutter was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Participants with known history of atrial fibrillation or atrial flutter were included and electrocardiogram confirmation was not required. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.60 | 0.48
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.074, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.98 to 1.6]

42. Secondary Outcome: Base Study: Time to First All-Cause Death Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated all-cause death was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. The analysis includes data obtained from vital status data collections of participants no longer followed in the base study. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.55 | 1.38
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.127, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.97 to 1.29]

43. Secondary Outcome: Base Study: Time to First Cardiovascular Death Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated cardiovascular death was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. The analysis includes data obtained from vital status data collections of participants no longer followed in the base study. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.45 | 0.39
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.277, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.89 to 1.52]

44. Secondary Outcome: Base Study: Time to First Fatal or Non-Fatal Myocardial Infarction Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal or non-fatal definite myocardial infarction was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.25 | 0.31
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.256, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.58 to 1.15]

45. Secondary Outcome: Base Study: Time to First Fatal Myocardial Infarction Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal definite myocardial infarction was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.03 | 0.03
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.794, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.29 to 2.57]

46. Secondary Outcome: Base Study: Time to First Fatal or Non-Fatal Stroke Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal or non-fatal definite stroke was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.58 | 0.44
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.034, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.02 to 1.7]

47. Secondary Outcome: Base Study: Time to First Fatal Stroke Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal definite stroke was determined for the base study using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.09 | 0.05
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.081, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.91, 95% CI 2-sided [0.93 to 3.97]

48. Secondary Outcome: Base Study + First Extension: Percent Change From Baseline in BMD Measurements of the Femoral Neck
Description: BMD was measured by DXA for all participants at the femoral neck-hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study + first extension-dbp).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 74 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (femoral neck BMD) was used for analysis (base study + first extension-dbp).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6498 | 6601
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 2.17 [1.78 to 2.55] | 0.70 [0.32 to 1.08]
  Month 12 | 2.81 [2.70 to 2.92] | 0.60 [0.49 to 0.71]
  Month 24: number analyzed (Participants) | 5924 | 5899
  Month 24 | 4.03 [3.90 to 4.16] | -0.36 [-0.49 to -0.22]
  Month 36: number analyzed (Participants) | 5294 | 5069
  Month 36 | 5.48 [5.32 to 5.64] | -1.02 [-1.18 to -0.86]
  Month 48: number analyzed (Participants) | 3807 | 3338
  Month 48 | 6.37 [6.17 to 6.56] | -1.93 [-2.13 to -1.73]
  Month 60: number analyzed (Participants) | 3181 | 2599
  Month 60 | 7.30 [7.08 to 7.53] | -2.75 [-2.99 to -2.51]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.47, 95% CI 2-sided [0.92 to 2.01]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.21, 95% CI 2-sided [2.05 to 2.37]
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.39, 95% CI 2-sided [4.20 to 4.57]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.50, 95% CI 2-sided [6.28 to 6.72]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.29, 95% CI 2-sided [8.02 to 8.57]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 10.05, 95% CI 2-sided [9.72 to 10.38]

49. Secondary Outcome: Base Study + First Extension: Percent Change From Baseline in BMD Measurements of the Distal-Third Forearm
Description: BMD was measured by DXA at the distal one-third radius at randomization and at yearly intervals until the end of the study (base study + first extension-dbp) in an approximate 10% random subset of participants at selected sites.
Time Frame: Baseline and once yearly, up to approximately 74 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (distal one-third radius BMD) was used for analysis (base study + first extension-dbp).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 679 | 718
Percent change
  Month 12 | 0.50 [0.18 to 0.81] | -0.61 [-0.91 to -0.30]
  Month 24: number analyzed (Participants) | 619 | 634
  Month 24 | 0.33 [-0.01 to 0.68] | -1.02 [-1.37 to -0.68]
  Month 36: number analyzed (Participants) | 576 | 564
  Month 36 | 0.05 [-0.33 to 0.43] | -1.91 [-2.29 to -1.53]
  Month 48: number analyzed (Participants) | 251 | 217
  Month 48 | -0.30 [-0.84 to 0.23] | -2.49 [-3.05 to -1.92]
  Month 60: number analyzed (Participants) | 328 | 263
  Month 60 | -0.84 [-1.37 to -0.31] | -3.17 [-3.74 to -2.59]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.10, 95% CI 2-sided [0.66 to 1.54]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.36, 95% CI 2-sided [0.87 to 1.85]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.96, 95% CI 2-sided [1.42 to 2.50]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.18, 95% CI 2-sided [1.40 to 2.96]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p = 0.001, Longitudinal model; Difference in Least Squares Means = 2.33, 95% CI 2-sided [1.54 to 3.11]

50. Secondary Outcome: Base Study + First Extension: Time From Baseline to First Osteoporotic Clinical Vertebral Fracture (Adjudicated)
Description: as for outcome 19
Time Frame: Up to approximately 74 months of observation
Population: The FAS including all randomized participants who took at least one dose of study medication with follow-up from start of prime therapy to study termination (base study + first extension) was used for analysis.
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.18 | 0.56
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.24 to 0.45]

51. Secondary Outcome: Base Study + First Extension: Time From Baseline to First Osteoporotic Clinical Fracture (Adjudicated)
Description: Osteoporotic clinical fractures (combining vertebral and non-vertebral) were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Vertebral fractures were assessed for all vertebral levels (C7, T1 to T12, L1 to L5). Non-vertebral fractures were assessed across multiple anatomical sites including clavicle, distal femur or shaft, fibula, hip, humerus, pelvis, radius, ribs, sacrum, tibia, ulna, and wrist. Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence rate of participants with fracture (number of participants with a fracture per 100 person-years of follow-up) is provided.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 50
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.95 | 2.93
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.60 to 0.75]

52. Secondary Outcome: Base Study + First Extension: Percent Change From Baseline in BMD Measurements of the Total Hip
Description: BMD was measured by DXA for all participants at the total hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study + first extension-dbp).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 74 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (total hip BMD) was used for analysis (base study + first extension-dbp).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6498 | 6601
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 1.89 [1.60 to 2.17] | 0.55 [0.26 to 0.83]
  Month 12 | 2.84 [2.75 to 2.92] | 0.34 [0.26 to 0.43]
  Month 24: number analyzed (Participants) | 5924 | 5899
  Month 24 | 3.79 [3.68 to 3.90] | -0.67 [-0.78 to -0.57]
  Month 36: number analyzed (Participants) | 5294 | 5069
  Month 36 | 4.78 [4.65 to 4.92] | -1.67 [-1.81 to -1.54]
  Month 48: number analyzed (Participants) | 3806 | 3338
  Month 48 | 5.52 [5.35 to 5.69] | -2.97 [-3.14 to -2.79]
  Month 60: number analyzed (Participants) | 3180 | 2599
  Month 60 | 6.23 [6.02 to 6.44] | -4.06 [-4.28 to -3.84]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.34, 95% CI 2-sided [0.94 to 1.74]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.50, 95% CI 2-sided [2.38 to 2.62]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.47, 95% CI 2-sided [4.31 to 4.62]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 6.46, 95% CI 2-sided [6.26 to 6.65]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.48, 95% CI 2-sided [8.24 to 8.73]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 10.29, 95% CI 2-sided [9.99 to 10.59]

53. Secondary Outcome: Base Study + First Extension: Percent Change From Baseline in BMD Measurements of the Trochanter
Description: BMD was measured by DXA for all participants at the trochanter-hip at screening, Months 6, 12, and subsequent yearly intervals until the end of the study (base study + first extension-dbp).
Time Frame: Baseline, Month 6, and once yearly, up to approximately 74 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (trochanter BMD) was used for analysis (base study + first extension-dbp).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6498 | 6601
Percent change
  Month 6: number analyzed (Participants) | 292 | 302
  Month 6 | 2.70 [2.21 to 3.18] | 0.95 [0.47 to 1.43]
  Month 12 | 4.33 [4.19 to 4.47] | 0.83 [0.69 to 0.97]
  Month 24: number analyzed (Participants) | 5924 | 5899
  Month 24 | 6.17 [6.00 to 6.34] | -0.23 [-0.40 to -0.06]
  Month 36: number analyzed (Participants) | 5294 | 5069
  Month 36 | 7.96 [7.75 to 8.16] | -1.29 [-1.50 to -1.08]
  Month 48: number analyzed (Participants) | 3806 | 3338
  Month 48 | 9.27 [9.01 to 9.53] | -2.86 [-3.13 to -2.59]
  Month 60: number analyzed (Participants) | 3180 | 2599
  Month 60 | 10.66 [10.36 to 10.97] | -3.90 [-4.22 to -3.57]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 1.74, 95% CI 2-sided [1.06 to 2.42]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 3.50, 95% CI 2-sided [3.31 to 3.70]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo at Month 24; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 6.41, 95% CI 2-sided [6.16 to 6.65]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.25, 95% CI 2-sided [8.95 to 9.54]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 12.14, 95% CI 2-sided [11.76 to 12.51]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 6]; Test type: Other; p < 0.001, Longitudinal model; [statistical method as in outcome 25, analysis 3]; Difference in Least Squares Means = 14.56, 95% CI 2-sided [14.11 to 15.01]

54. Secondary Outcome: Base Study + First Extension: Percent Change From Baseline in BMD Measurements of the Lumbar Spine
Description: BMD was measured by DXA for all participants at the lumbar spine at randomization, Months 6, 12, and subsequent yearly intervals until the end of the study (base study + first extension-dbp). Measurements were made on at least 3 vertebrae for all time points; vertebrae with fractures were excluded from analyses.
Time Frame: Baseline, Month 6, and once yearly, up to approximately 74 months of observation
Population: The FAS population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (lumbar spine BMD) was used for analysis (base study + first extension-dbp).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 6220 | 6375
Percent change
  Month 6: number analyzed (Participants) | 291 | 298
  Month 6 | 3.72 [3.36 to 4.07] | 0.82 [0.47 to 1.17]
  Month 12 | 4.61 [4.50 to 4.71] | 0.60 [0.49 to 0.70]
  Month 24: number analyzed (Participants) | 5682 | 5753
  Month 24 | 6.63 [6.50 to 6.76] | 0.70 [0.58 to 0.83]
  Month 36: number analyzed (Participants) | 5682 | 5753
  Month 36 | 8.41 [8.26 to 8.56] | 0.72 [0.56 to 0.87]
  Month 48: number analyzed (Participants) | 5105 | 5008
  Month 48 | 10.19 [10.01 to 10.38] | 0.85 [0.66 to 1.04]
  Month 60: number analyzed (Participants) | 3066 | 2547
  Month 60 | 11.93 [11.71 to 12.15] | 1.06 [0.83 to 1.29]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.90, 95% CI 2-sided [2.40 to 3.39]
Statistical Analysis 2: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 2]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 4.01, 95% CI 2-sided [3.87 to 4.15]
Statistical Analysis 3: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 3]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 5.93, 95% CI 2-sided [5.75 to 6.11]
Statistical Analysis 4: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 7.70, 95% CI 2-sided [7.48 to 7.91]
Statistical Analysis 5: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.34, 95% CI 2-sided [9.08 to 9.61]
Statistical Analysis 6: Comparison: Odanacatib 50 mg OW vs Placebo; [analysis description as in outcome 22, analysis 5]; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 10.87, 95% CI 2-sided [10.55 to 11.19]

55. Secondary Outcome: Base Study + First Extension + Second Extension: Time From Baseline to First Morphometrically-Assessed Vertebral Fracture
Description: Morphometric vertebral fractures were assessed by central adjudication on lumbar and thoracic spinal radiographs acquired at baseline (base study) and at Months 6, 12, and subsequent yearly time points. Incident fractures (i.e., occurring after baseline) in previously normal vertebral bodies and/or those occurring after baseline in previously fractured vertebral bodies (Genant semiquantitative [SQ] Grade 1-3) (T4 to L4) were confirmed by quantitative morphometric (QM) and either SQ or binary SQ (yes/no) methodologies. A time-to-event methodology was used to evaluate results: life-table estimates of the incidence proportion (cumulative incidence) of participants with at least one morphometric vertebral fracture were assessed at Months 6, 12, and subsequent yearly intervals; an interval-censored approach was then used to determine incidence rate (number of participants with a morphometric fracture per 100 person-years of follow-up).
Time Frame: Up to approximately 108 months of observation
Population: Study was terminated early due to observed increase in risk of stroke in Protocol MK-0822-018. As a result, efficacy analyses in 2nd Extension were limited to change in BMD and incidence of osteoporotic clinical fractures; Base Study + 1st Ext + 2nd Ext: Time From Baseline to First Morphometrically-Assessed Vertebral Fracture was not analyzed.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Base Study + First Extension + Second Extension: Change in Height From Baseline Stature
Description: Height was measured by wall-mounted stadiometer at randomization and at yearly intervals across the base study and the two extension studies.
Time Frame: Baseline and once yearly, up to approximately 108 months of observation
Population: Study was terminated early due to observed increase in risk of stroke in Protocol MK-0822-018. As a result, efficacy analyses in 2nd Extension were limited to change in BMD and incidence of osteoporotic clinical fractures; Base Study + First Extension + Second Extension: Change in Height from Baseline Stature was not analyzed.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Base Study + First Extension + Second Extension: Percent Change From Baseline in BMD Measurements of the Lumbar Spine
Description: BMD was measured by DXA at the lumbar spine starting at randomization, and at yearly intervals until the end of the study (2nd extension study) for all participants who entered the 2nd extension study. Measurements were made on at least 3 vertebrae for all time points; vertebrae with fractures were excluded from analyses. At Months 96 and 108, approximately 3% or fewer participants in each treatment group had BMD data, and results at those time points should be viewed with caution. NOTE: The mean percent change in BMD from baseline in participants originally randomized to placebo includes BMD results obtained after those participants were switched to open-label odanacatib, which occurred at different times relative to their start of blinded study medication in the base study. A longitudinal model with terms for treatment, stratum, region & interaction between treatment and time as fixed effects (LS means weighted for region & stratum size) was used for analysis.
Time Frame: Baseline and once yearly, up to approximately 108 months of observation
Population: The FAS population consisted of all randomized participants who entered the second extension study and received at least one dose of open-label treatment and had the necessary on-treatment information (lumbar spine BMD).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 2818 | 2128
Percent change
  Month 12 | 4.68 [4.54 to 4.83] | 1.01 [0.84 to 1.17]
  Month 24: number analyzed (Participants) | 2803 | 2121
  Month 24 | 6.95 [6.78 to 7.12] | 1.40 [1.21 to 1.59]
  Month 36: number analyzed (Participants) | 2798 | 2117
  Month 36 | 8.84 [8.65 to 9.04] | 1.61 [1.39 to 1.83]
  Month 48: number analyzed (Participants) | 2754 | 2077
  Month 48 | 10.74 [10.51 to 10.97] | 2.06 [1.80 to 2.33]
  Month 60: number analyzed (Participants) | 2604 | 1975
  Month 60 | 12.55 [12.29 to 12.81] | 2.45 [2.16 to 2.75]
  Month 72: number analyzed (Participants) | 2068 | 1594
  Month 72 | 13.76 [13.46 to 14.06] | 6.25 [5.91 to 6.59]
  Month 84: number analyzed (Participants) | 1538 | 1152
  Month 84 | 14.91 [14.56 to 15.26] | 8.37 [7.97 to 8.77]
  Month 96: number analyzed (Participants) | 208 | 177
  Month 96 | 15.13 [14.48 to 15.78] | 9.66 [8.95 to 10.38]
  Month 108: number analyzed (Participants) | 56 | 47
  Month 108 | 15.54 [14.23 to 26.85] | 10.85 [9.42 to 12.27]

58. Secondary Outcome: Base Study + First Extension + Second Extension: Percent Change From Baseline in BMD Measurements of the Femoral Neck
Description: BMD was measured by DXA at the femoral neck starting at screening, and at yearly intervals until the end of the study (2nd extension study) for all participants who entered the 2nd extension study. LS means percent change in BMD from original baseline are provided through Month 108. At Months 96 and 108, approximately 3% or fewer participants in each treatment group had BMD data, and results at those time points should be viewed with caution. NOTE: The mean percent change in BMD from baseline in participants originally randomized to placebo includes BMD results obtained after those participants were switched to open-label odanacatib, which occurred at different times relative to their start of blinded study medication in the base study. A longitudinal model with terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS means weighted for region and stratum size) was used for analysis.
Time Frame: Baseline and once yearly, up to approximately 108 months of observation
Population: The FAS population consisted of all randomized participants who entered the second extension study and received at least one dose of open-label treatment and had the necessary on-treatment information (femoral neck BMD).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 2997 | 2212
Percent change
  Month 12 | 2.89 [2.73 to 3.05] | 1.06 [0.88 to 1.24]
  Month 24: number analyzed (Participants) | 2965 | 2189
  Month 24 | 4.39 [4.20 to 4.57] | 0.38 [0.17 to 0.60]
  Month 36: number analyzed (Participants) | 2950 | 2171
  Month 36 | 6.02 [5.81 to 6.24] | -0.03 [-0.28 to 0.22]
  Month 48: number analyzed (Participants) | 2905 | 2133
  Month 48 | 7.01 [6.78 to 7.25] | -0.73 [-1.01 to -0.46]
  Month 60: number analyzed (Participants) | 2718 | 2015
  Month 60 | 7.98 [7.70 to 8.25] | -1.32 [-1.63 to -1.00]
  Month 72: number analyzed (Participants) | 2186 | 1637
  Month 72 | 8.51 [8.21 to 8.81] | 0.41 [0.06 to 0.76]
  Month 84: number analyzed (Participants) | 1631 | 1197
  Month 84 | 9.11 [8.75 to 9.48] | 1.56 [1.13 to 1.98]
  Month 96: number analyzed (Participants) | 237 | 187
  Month 96 | 8.84 [8.22 to 9.46] | 1.95 [1.24 to 2.65]
  Month 108: number analyzed (Participants) | 63 | 51
  Month 108 | 9.38 [7.83 to 10.92] | 3.63 [1.91 to 5.35]

59. Secondary Outcome: Base Study + First Extension + Second Extension: Percent Change From Baseline in BMD Measurements of the Trochanter
Description: BMD was measured by DXA at the trochanter starting at screening, and at yearly intervals until the end of the study (2nd extension study) for all participants who entered the 2nd extension study. LS means percent change in BMD from original baseline are provided through Month 108. At Months 96 and 108, approximately 3% or fewer participants in each treatment group had BMD data, and results at those time points should be viewed with caution. NOTE: The mean percent change in BMD from baseline in participants originally randomized to placebo includes BMD results obtained after those participants were switched to open-label odanacatib, which occurred at different times relative to their start of blinded study medication in the base study. A longitudinal model with terms for treatment, stratum, region and interaction between treatment and time as fixed effects (LS means weighted for region and stratum size) was used for analysis.
Time Frame: Baseline and once yearly, up to approximately 108 months of observation
Population: The FAS population consisted of all randomized participants who entered the second extension study and received at least one dose of open-label treatment and had the necessary on-treatment information (trochanter BMD).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 2997 | 2212
Percent change
  Month 12 | 4.55 [4.34 to 4.75] | 1.81 [1.58 to 2.05]
  Month 24: number analyzed (Participants) | 2965 | 2171
  Month 24 | 6.85 [6.62 to 7.08] | 1.45 [1.18 to 1.72]
  Month 36: number analyzed (Participants) | 2950 | 2171
  Month 36 | 9.00 [8.73 to 9.28] | 0.89 [0.57 to 1.21]
  Month 48: number analyzed (Participants) | 2905 | 2171
  Month 48 | 10.58 [10.26 to 10.89] | -0.16 [-0.52 to 0.21]
  Month 60: number analyzed (Participants) | 2718 | 2133
  Month 60 | 12.21 [11.85 to 12.57] | -0.68 [-1.09 to -0.26]
  Month 72: number analyzed (Participants) | 2186 | 1637
  Month 72 | 12.95 [12.55 to 13.34] | 1.22 [0.76 to 1.68]
  Month 84: number analyzed (Participants) | 1631 | 1197
  Month 84 | 13.30 [12.82 to 13.78] | 3.17 [2.61 to 3.73]
  Month 96: number analyzed (Participants) | 237 | 187
  Month 96 | 13.44 [12.67 to 14.20] | 4.66 [3.79 to 5.54]
  Month 108: number analyzed (Participants) | 63 | 51
  Month 108 | 12.69 [10.86 to 14.51] | 2.97 [0.95 to 5.00]

60. Secondary Outcome: Second Extension: Incidence of Osteoporotic Clinical Lumbar Vertebral Fracture (Adjudicated)
Description: Osteoporotic vertebral clinical fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Vertebral fractures were assessed for all lumbar vertebral levels (L1 to L5). Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence of participants in the second extension study with osteoporotic vertebral clinical fractures is provided. Due to early termination of the study, the cumulative incidence using a time-to-event methodology was not assessed across base and extension studies.
Time Frame: Up to approximately 34 months of observation
Population: The All-Participants-as-Treated Population including all randomized participants who entered the second extension study and received at least one dose of open-label treatment was used for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 3114 | 2309
Percentage of Participants | 0.22 | 0.04

61. Secondary Outcome: Second Extension: Incidence of Osteoporotic Clinical Thoracic Vertebral Fracture (Adjudicated)
Description: Osteoporotic vertebral clinical fractures were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Vertebral fractures were assessed for all thoracic vertebral levels (T1 to T12). Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence of participants in the second extension study with osteoporotic vertebral clinical fractures is provided. Due to early termination of the study, the cumulative incidence using a time-to-event methodology was not assessed across base and extension studies.
Time Frame: Up to approximately 34 months of observation
Population: as for outcome 60
Measure: Number; unit: Percentage of Participants
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 3114 | 2309
Percentage of Participants | 0.13 | 0.09

62. Secondary Outcome: Second Extension: Time From Baseline to First Osteoporotic Clinical Fracture of Any Type (Adjudicated)
Description: Osteoporotic clinical fractures of any type were confirmed by central adjudication using radiographic evidence on all symptomatic fractures reported as adverse experiences (excluding fractures of the fingers, toes, face, and skull). Non-vertebral fractures were assessed across multiple anatomical sites including clavicle, distal femur or shaft, fibula, hip, humerus, pelvis, radius, ribs, sacrum, tibia, ulna, and wrist; Vertebral fractures assessed across all vertebral levels (C7, T1 to T12, L1 to L5) were included in the analysis. Osteoporotic (fragility) fractures did not include fractures with traumatic or pathological etiologies. A clinical fracture was defined as a fracture with clinical fracture-related symptoms (e.g., pain). A time-to-event methodology was used to evaluate results: the incidence proportion (cumulative incidence) of participants in the second extension study with at least one osteoporotic clinical fracture of any type is provided.
Time Frame: Up to approximately 34 months of observation
Population: The The All-Participants-as-Treated Population including all randomized participants who entered the second extension study and received at least one dose of open-label treatment was used for analysis.
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 3144 | 2309
Parts. with event per 100 person-years | 2.04 | 2.64

63. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in Cortical vBMD of the Total Hip Using Quantitative Computed Tomography
Description: Compartment-specific effects of osteoporosis were assessed by measuring cortical vBMD at the total hip using quantitative computed tomography. The percent change from baseline at Month 24 was then assessed using a longitudinal data analysis model including terms for treatment, stratum (prior vertebral fracture [yes/no]) and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (total hip cortical vBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 51 | 55
Percent change | 3.29 [2.33 to 4.24] | 0.52 [-0.39 to 1.44]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 2.76, 95% CI 2-sided [1.43 to 4.10]

64. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in Areal BMD (aBMD) of the Lumbar Spine Using DXA
Description: aBMD was measured at the lumbar spine (L1 to L4) at baseline and Month 24 using DXA . If a vertebra was fractured at baseline or became fractured during the study, its BMD measurement was excluded from analysis. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (lumbar spine aBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 50 | 59
Percent change | 5.63 [4.54 to 6.72] | 0.08 [-0.92 to 1.09]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 5.55, 95% CI 2-sided [4.06 to 7.05]

65. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in aBMD of the Femoral Neck Using DXA
Description: aBMD was measured at the femoral neck at baseline and Month 24 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (femoral neck aBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 49 | 58
Percent change | 3.15 [1.74 to 4.56] | 0.36 [-0.94 to 1.65]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.005, Longitudinal model; Difference in Least Squares Means = 2.79, 95% CI 2-sided [0.86 to 4.72]

66. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in aBMD of the Total Hip Using DXA
Description: aBMD was measured at the total hip at baseline and Month 24 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (total hip aBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 49 | 58
Percent change | 2.96 [2.03 to 3.90] | -0.66 [-1.52 to 0.20]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 3.63, 95% CI 2-sided [2.35 to 4.90]

67. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in aBMD of the Trochanter Using DXA
Description: aBMD was measured at the trochanter at baseline and Month 24 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (trochanter aBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 49 | 58
Percent change | 5.10 [3.74 to 6.45] | -0.55 [-1.80 to 0.70]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 5.65, 95% CI 2-sided [3.79 to 7.50]

68. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in s-CTx After Log-Transformation
Description: s-CTx, a biochemical marker of bone resorption by osteoclasts reflecting collagen breakdown products, was assessed at baseline and Month 24 in an approximate 10% random subset participants at selected sites in the P018 base study who were additionally included in the imaging substudy PN032-base study. The log-transformed fraction from baseline in s-CTx was determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 24
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (s-CTx) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (PN032-Base).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 45
Percent change | -55.62 [-62.53 to -47.44] | 6.62 [-8.51 to 24.26]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -62.25, 95% CI 2-sided [-79.99 to -44.50]

69. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in P1NP After Log-Transformation
Description: P1NP is a cleavage fragment produced during the synthesis of collagenous bone matrix (type 1 collagen) used as a biochemical marker of bone formation. Serum P1NP was assessed at baseline and Month 24 in an approximate 10% random subset participants at selected sites in the P018 base study who were additionally included in the imaging substudy PN032-base study. The log-transformed fraction change from baseline in P1NP was determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 24
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (P1NP) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (PN032-Base).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 45
Percent change | -33.56 [-42.66 to -23.01] | -6.86 [-18.71 to 6.72]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.001, Longitudinal model; Difference in Least Squares Means = -26.70, 95% CI 2-sided [-42.56 to -10.83]

70. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in aBMD of the Distal-Third Forearm Using DXA
Description: aBMD was measured at the the distal one-third radius at baseline and Month 24 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 24
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (distal one-third radius aBMD) was used for analysis (PN032-Base).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 49 | 55
Percent change | 0.40 [-0.57 to 1.36] | -1.27 [-2.18 to -0.36]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.016, Longitudinal model; Difference in Least Squares Means = 1.67, 95% CI 2-sided [0.32 to 3.01]

71. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in BSAP After Log-Transformation
Description: BSAP is an enzyme produced by matrix-synthesizing osteoblasts during the synthesis of collagenous bone matrix (type 1 collagen) used as a biochemical marker of bone formation. Serum BSAP was assessed at baseline and Month 24 in an approximate 10% random subset participants at selected sites in the P018 base study who were additionally included in the imaging substudy PN032-base study. The log-transformed fraction from baseline in BSAP was determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 24
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (BSAP) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (PN032-Base).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 45
Percent change | -12.39 [-19.20 to -4.99] | 12.64 [4.53 to 21.38]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -25.02, 95% CI 2-sided [-35.92 to -14.12]

72. Secondary Outcome: Imaging Substudy PN032-Base: Percent Change From Baseline in u-NTx/Cr Ratio After Log-Transformation
Description: u-NTx, a biochemical marker of bone resorption by osteoclasts reflecting collagen breakdown products, was assessed at baseline and Month 24 in an approximate 10% random subset participants at selected sites in the P018 base study who were additionally included in the imaging substudy PN032-base study. Urine NTx measurements (in BCE) were normalized to urine Cr concentration (i.e., u-NTx/Cr ratio) and the log-transformed fraction from baseline in u-NTx/Cr ratio was then determined using a longitudinal model with terms for treatment, stratum, and interaction between treatment and time as fixed effects (LS means weighted for stratum size). Back-transformed weighted geometric LS means values for percent change from baseline are provided.
Time Frame: Baseline, Month 24
Population: The per-protocol population including all randomized participants who took at least one dose of study medication and having the necessary on-treatment information (u-NTx/Cr) and excluding participants and/or data points that represent clinically important deviations from the protocol-specified criteria was used for analysis (PN032-Base).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo: Participants received blinded placebo to 50 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). This was to be followed by 50 mg of open-label odanacatib weekly for 5 up to years. Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 45
Percent change | -47.87 [-57.26 to -36.42] | 16.56 [-2.85 to 39.84]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = -64.43, 95% CI 2-sided [-87.80 to -41.07]

73. Secondary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in Cortical vBMD of the Total Hip Using Quantitative Computed Tomography
Description: Compartment-specific effects of osteoporosis were assessed by measuring cortical vBMD at the total hip using quantitative computed tomography. The percent change from baseline at Month 60 (base study + extension study) was then assessed using a longitudinal data analysis model including terms for treatment, stratum (prior vertebral fracture [yes/no]) and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: as for outcome 63
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 32 | 27
Percent change | 6.00 [4.07 to 7.93] | -2.53 [-4.48 to -0.59]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 8.53, 95% CI 2-sided [5.79 to 11.28]

74. Secondary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in aBMD of the Lumbar Spine Using DXA
Description: aBMD was measured at the lumbar spine (L1 to L4) at baseline and Month 60 using DXA . If a vertebra was fractured at baseline or became fractured during the study, its BMD measurement was excluded from analysis. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (lumbar spine aBMD) was used for analysis (PN032-Base + Extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 37
Percent change | 11.80 [9.86 to 13.73] | 0.72 [-1.10 to 2.54]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 11.08, 95% CI 2-sided [8.41 to 13.74]

75. Secondary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in aBMD of the Total Hip Using DXA
Description: aBMD was measured at the total hip at baseline and Month 60 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (total hip aBMD) was used for analysis (PN032-Base + Extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 38 | 35
Percent change | 5.34 [3.66 to 7.01] | -5.07 [-6.74 to -3.41]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 10.41, 95% CI 2-sided [8.05 to 12.78]

76. Secondary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in aBMD of the Femoral Neck Using DXA
Description: aBMD was measured at the femoral neck at baseline and Month 60 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (femoral neck aBMD) was used for analysis (PN032-Base + Extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 38 | 35
Percent change | 6.87 [4.68 to 9.06] | -3.11 [-5.26 to -0.96]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 9.98, 95% CI 2-sided [6.91 to 13.06]

77. Secondary Outcome: Imaging Substudy PN032-Base + Extension: Percent Change From Baseline in aBMD of the Trochanter Using DXA
Description: aBMD was measured at the trochanter at baseline and Month 60 using DXA. The percent change from baseline was assessed using a longitudinal data analysis model including terms for treatment, stratum and interaction between treatment and time as fixed effects (LS means weighted for stratum size).
Time Frame: Baseline, Month 60
Population: The FAS including consisting of all randomized participants who took at least one dose of blinded study treatment and have a baseline and at least one on-treatment measurement available (trochanter aBMD) was used for analysis (PN032-Base + Extension).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 36 | 37
Percent change | 10.44 [7.84 to 13.03] | -4.50 [-7.07 to -1.94]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p < 0.001, Longitudinal model; Difference in Least Squares Means = 14.94, 95% CI 2-sided [11.29 to 18.59]

78. Other Pre Specified Outcome: Base Study + First Extension: Time to First Hospitalization for Unstable Angina Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated hospitalization for unstable angina was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.08 | 0.10
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.366, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.47 to 1.33]

79. Other Pre Specified Outcome: Base Study + First Extension: Time to First Cardiovascular Death Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated cardiovascular death was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. The analysis includes data obtained from vital status data collections of participants no longer followed in the base study. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.48 | 0.43
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.246, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.92 to 1.4]

80. Other Pre Specified Outcome: Base Study + First Extension: Time to First Fatal Myocardial Infarction Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal definite myocardial infarction was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.02 | 0.03
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.638, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.32 to 2.03]

81. Other Pre Specified Outcome: Base Study + First Extension: Time to First 3-Point MACE Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated 3-point MACE (a composite outcome measure of 1. cardiovascular death, 2. non-fatal definite MI, or 3. non-fatal definite stroke) was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.24 | 1.06
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.029, Regression, Cox; No adjustments for multiplicity were applied; p-value is unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.02 to 1.36]

82. Other Pre Specified Outcome: Base Study + First Extension: Time to First All-Cause Death Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated all-cause death was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. The analysis includes data obtained from vital status data collections of participants no longer followed in the base study. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.79 | 1.70
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.341, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.95 to 1.17]

83. Other Pre Specified Outcome: Base Study + First Extension: Time to First New Onset ECG-Confirmed Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated new or presumed new onset atrial fibrillation or atrial flutter was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Participants with known history of atrial fibrillation or atrial flutter were excluded and electrocardiogram confirmation was required. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.27 | 0.22
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.198, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.9 to 1.68]

84. Other Pre Specified Outcome: Base Study + First Extension: Time to First Fatal or Non-Fatal Myocardial Infarction Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal or non-fatal definite myocardial infarction was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.26 | 0.28
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.798, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.7 to 1.26]

85. Other Pre Specified Outcome: Base Study + First Extension: Time to First Fatal or Non-Fatal Stroke Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal or non-fatal definite stroke was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.58 | 0.42
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.005, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [1.1 to 1.71]

86. Other Pre Specified Outcome: Base Study + First Extension: Time to First Any Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: as for outcome 41
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.61 | 0.50
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.059, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.99 to 1.5]

87. Other Pre Specified Outcome: Base Study + First Extension: Time to First Fatal Stroke Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated fatal definite stroke was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.09 | 0.05
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.114, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [0.89 to 2.9]

88. Other Pre Specified Outcome: Base Study + First Extension: Time to First 4-Point MACE Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated 4-point MACE (a composite outcome measure of 1. cardiovascular death, 2. non-fatal definite MI, 3. non-fatal definite stroke, or 4. hospitalization for unstable angina) was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 1.31 | 1.15
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.159, Regression, Cox; No adjustments for multiplicity were applied; p-value is unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.99 to 1.31]

89. Other Pre Specified Outcome: Base Study + First Extension: Time to First New Onset Atrial Fibrillation or Atrial Flutter Confirmed by TIMI Adjudication
Description: The time to first TIMI-adjudicated new or presumed new onset atrial fibrillation or atrial flutter was determined for the base study + first extension using a Cox proportional hazards model with terms for treatment, stratum and geographic region. Participants with known history of atrial fibrillation or atrial flutter were excluded and electrocardiogram confirmation was not required. Results are expressed as number of participants with an event per 100 person-years of follow-up. Results from MK-0822-083, a follow up study to the MK-088-018 base study and the double-blind period of the first extension study for participants who discontinued prior to 5 years follow-up, are not included.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number; unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.51 | 0.43
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Odanacatib 50 mg OW - Placebo; Test type: Other; p = 0.178, Regression, Cox; No adjustments for multiplicity were applied; all p-values reported were unadjusted and therefore considered nominal; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.93 to 1.46]

90. Post Hoc Outcome: Base Study: Incidence Rate of Femoral Shaft Fractures Confirmed by Adjudication
Description: The incidence rate of femoral shaft fracture events (including both atypical and non-atypical; of any etiology including traumatic) confirmed by adjudication was determined for the base study. Results are expressed as number of participants with an event per 100 person-years of follow-up.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.10 [0.06 to 0.15] | 0.06 [0.03 to 0.10]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.04, 95% CI 2-sided [-0.01 to 0.09]

91. Post Hoc Outcome: Base Study: Incidence Rate of Atypical Femoral Shaft Fractures Confirmed by Adjudication
Description: Atypical subtrochanteric/diaphyseal femoral fractures (AFF) are an uncommon type of low-energy (eg, osteoporotic) femoral shaft fracture of unclear causation infrequently reported in osteoporotic persons treated with long-term anti-resorptive therapy (eg, bisphosphonates). All femoral (femur, femur-distal, femur-shaft) fractures in the base study were adjudicated against both ASBMR 2010 and 2013 criteria. All 5 major features (ie, location along femoral shaft, no/minimal trauma, transverse/short oblique fracture, non-comminuted, complete/incomplete fracture) were required for ASBMR 2010 AFF case definition; while 4 of 5 major features (ie, no/minimal trauma, substantially transverse orientation at cortical origin with possible oblique orientation medially, non-comminuted/minimally comminuted, complete/incomplete fracture, localized periosteal reaction of lateral cortex) with requirement for location along femoral shaft were required for ASBMR 2013 AFF case definition.
Time Frame: Up to approximately 60 months of observation
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.02 [0.01 to 0.05] | 0.00 [0.00 to 0.02]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.02, 95% CI 2-sided [0.01 to 0.05]

92. Post Hoc Outcome: Base Study + First Extension: Incidence Rate of Femoral Shaft Fractures Confirmed by Adjudication
Description: The incidence rate of femoral shaft fracture events (including both atypical and non-atypical; of any etiology including traumatic) confirmed by adjudication was determined for the base study + first extension. Results are expressed as number of participants with an event per 100 person-years of follow-up.
Time Frame: Up to approximately 74 months of observation
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.09 [0.06 to 0.13] | 0.02 [0.01 to 0.05]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.06, 95% CI 2-sided [0.03 to 0.11]

93. Post Hoc Outcome: Base Study + First Extension: Incidence Rate of Atypical Femoral Shaft Fractures Confirmed by Adjudication
Description: Atypical subtrochanteric/diaphyseal femoral fractures (AFF) are an uncommon type of low-energy (eg, osteoporotic) femoral shaft fracture of unclear causation infrequently reported in osteoporotic persons treated with long-term anti-resorptive therapy (eg, bisphosphonates). All femoral (femur, femur-distal, femur-shaft) fractures in the base study + first extension were adjudicated against both ASBMR 2010 & 2013 criteria. All 5 major features (ie, location along femoral shaft, no/minimal trauma, transverse/short oblique fracture, non-comminuted, complete/incomplete fracture) were required for ASBMR 2010 AFF case definition; while 4 of 5 major features (ie, no/minimal trauma, substantially transverse orientation at cortical origin with possible oblique orientation medially, non-comminuted/minimally comminuted, complete/incomplete fracture, localized periosteal reaction of lateral cortex) with requirement for location along femoral shaft were required for ASBMR 2013 AFF case definition.
Time Frame: Up to approximately 74 months of observation
Population: The All-Participants-as-Treated population, including all randomized participants who took at least one dose of study medication, was used for analysis (base study + first extension).
Measure: Number (95% Confidence Interval); unit: Parts. with event per 100 person-years
Arm/Group | Odanacatib 50 mg OW | Placebo
Number analyzed (Participants) | 8043 | 8028
Parts. with event per 100 person-years | 0.03 [0.02 to 0.06] | 0.00 [0.00 to 0.01]
Statistical Analysis 1: Comparison: Odanacatib 50 mg OW vs Placebo; Test type: Other — Miettinen & Nurminen; Difference in rates = 0.03, 95% CI 2-sided [0.02 to 0.06]

ADVERSE EVENTS:
Time Frame: Base Study + First Extension treatment groups: Up to approximately 74 months of observation Second Extension treatment groups: Up to approximately 34 months of observation
Description: The All-Participants-as-Treated population including all randomized patients who took at least one dose of study medication was used for analysis (base study + first extension; second extension).
Groups:
- Base Study + First Extension: Odanacatib 50 mg OW: Participants received 50 mg of blinded odanacatib weekly over the course of the base study and first extension study (5 years total). Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
- Base Study + First Extension: Placebo: Participants received blinded placebo to 10 mg of odanacatib weekly over the course of the base study and first extension study (5 years total). Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
- Second Extension: Odanacatib 50 mg OW: Participants received 50 mg of open-label odanacatib weekly for 5 years in the second extension study after having previously received 50 mg of blinded odanacatib weekly in the base study and first extension study (5 years total). Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
- Second Extension: Odanacatib 50 mg OW (Placebo): Participants received 50 mg of open-label odanacatib weekly for 5 years in the second extension study after having previously received blinded placebo to 50 mg of odanacatib weekly in the base study and first extension study (5 years total). Participants also received Vitamin D3 and open-label supplemental calcium so that total daily calcium intake (from both dietary and supplemental sources) was approximately 1200 mg.
Arm/Group | Base Study + First Extension: Odanacatib 50 mg OW | Base Study + First Extension: Placebo | Second Extension: Odanacatib 50 mg OW | Second Extension: Odanacatib 50 mg OW (Placebo)
All-Cause Mortality (participants affected / at risk) | 378/8043 | 327/8028 | 86/3144 | 39/2309
Serious Adverse Events (participants affected / at risk) | 2441/8043 | 2446/8028 | 508/3144 | 376/2309
Other Adverse Events (participants affected / at risk) | 5659/8043 | 5624/8028 | 311/3144 | 209/2309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study + First Extension: Odanacatib 50 mg OW (N=8043) | Base Study + First Extension: Placebo (N=8028) | Second Extension: Odanacatib 50 mg OW (N=3144) | Second Extension: Odanacatib 50 mg OW (Placebo) (N=2309)
Anaemia (Blood and lymphatic system disorders) | 16 (17) | 21 (22) | 4 (4) | 2 (2)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 17 (17) | 9 (9)
Acute myocardial infarction (Cardiac disorders) | 55 (57) | 55 (59) | 0 (0) | 0 (0)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 39 (44) | 41 (44) | 4 (4) | 2 (2)
Angina unstable (Cardiac disorders) | 34 (43) | 34 (37) | 4 (5) | 4 (4)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 5 (5) | 6 (7) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 73 (83) | 80 (97) | 17 (23) | 10 (10)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 6 (6) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 8 (9) | 6 (6) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 10 (10) | 6 (6) | 0 (0) | 0 (0)
Bundle branch block bilateral (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 10 (10) | 9 (10) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 9 (10) | 13 (13) | 2 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 35 (38) | 41 (44) | 7 (7) | 5 (6)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 7 (9) | 2 (5) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 37 (38) | 35 (36) | 10 (10) | 3 (5)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 11 (11) | 14 (14) | 4 (4) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 31 (34) | 25 (28) | 7 (7) | 6 (6)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cytotoxic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 47 (50) | 48 (51) | 4 (4) | 5 (5)
Myocardial ischaemia (Cardiac disorders) | 19 (21) | 12 (12) | 1 (1) | 6 (6)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Postinfarction angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 8 (8) | 9 (9) | 3 (3) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Congenital bronchiectasis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Exomphalos (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
External ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 15 (16) | 5 (5) | 3 (3) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 5 (6) | 2 (2) | 0 (0) | 1 (1)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Hyperadrenalism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 98 (131) | 79 (108) | 12 (16) | 9 (13)
Cataract nuclear (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choroiditis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Excessive eye blinking (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 8 (9) | 3 (4) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis interstitial (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lens disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Retinal dystrophy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Corneal scar (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flat anterior chamber of eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 9 (9) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 2 (2) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 7 (7) | 5 (5) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 8 (8) | 6 (6) | 0 (0) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 5 (5) | 7 (7) | 1 (1) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9) | 10 (10) | 2 (2) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 8 (9) | 2 (2) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 9 (9) | 9 (9) | 5 (6) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 7 (7) | 3 (4) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diverticulum oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dolichocolon acquired (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysbacteriosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 5 (6) | 7 (7) | 2 (2) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 19 (19) | 10 (11) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 7 (7) | 1 (1) | 3 (3)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 10 (10) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 11 (11) | 10 (10) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 7 (7) | 7 (8) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 7 (7) | 11 (11) | 1 (1) | 2 (2)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 11 (12) | 11 (12) | 3 (3) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Ischiorectal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 10 (10) | 2 (2) | 3 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (2) | 1 (1)
Lumbar hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Mesenteric artery embolism (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mouth cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 8 (8) | 6 (8) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 8 (8) | 5 (5) | 3 (3) | 2 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 2 (2)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 10 (10) | 2 (2) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (6) | 2 (2) | 1 (1)
Accidental death (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Adverse event (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 7 (8) | 3 (3) | 0 (0) | 0 (0)
Capsular contracture associated with breast implant (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 22 (23) | 24 (25) | 3 (4) | 4 (4)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 66 (66) | 62 (62) | 14 (14) | 4 (4)
Device adhesion issue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device damage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device material issue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Multi-organ disorder (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 10 (10) | 6 (6) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (5) | 6 (6) | 0 (0) | 4 (4)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Oral administration complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 7 (7) | 1 (1) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Strangulated hernia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 15 (15) | 2 (2) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 9 (10) | 3 (3) | 2 (2) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 20 (20) | 15 (15) | 3 (3) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 7 (7) | 15 (15) | 1 (1) | 3 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 34 (34) | 34 (38) | 7 (7) | 3 (3)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Amoebic colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 18 (18) | 12 (12) | 6 (6) | 3 (3)
Appendicitis perforated (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 15 (15) | 14 (15) | 4 (4) | 2 (2)
Bronchopneumonia (Infections and infestations) | 18 (19) | 17 (18) | 0 (0) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 15 (17) | 16 (20) | 3 (3) | 3 (3)
Central nervous system viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cutaneous tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 4 (4) | 8 (8) | 1 (1) | 0 (0)
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Dental fistula (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 25 (27) | 20 (22) | 4 (4) | 4 (4)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 6 (6) | 5 (7) | 0 (0) | 1 (1)
Erythema migrans (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 34 (34) | 26 (27) | 1 (1) | 3 (4)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bites (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected varicose vein (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 (5) | 7 (7) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal fistula infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 11 (11) | 12 (12) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 13 (13) | 9 (9) | 5 (6) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 4 (6) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 7 (7) | 5 (5) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 117 (134) | 116 (121) | 31 (32) | 19 (19)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (4) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary echinococciasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Pyelocystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 4 (4) | 7 (8) | 2 (3) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pyometra (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 23 (24) | 18 (19) | 2 (2) | 5 (5)
Septic shock (Infections and infestations) | 12 (12) | 7 (7) | 6 (6) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tick-borne fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 54 (58) | 49 (59) | 16 (16) | 9 (11)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Viral labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 7 (7) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 13 (15) | 19 (23) | 4 (4) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 5 (5) | 8 (8) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 6 (6) | 8 (8) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 15 (18) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 29 (29) | 62 (64) | 4 (4) | 9 (9)
Femur fracture (Injury, poisoning and procedural complications) | 44 (49) | 40 (41) | 8 (8) | 4 (5)
Fibula fracture (Injury, poisoning and procedural complications) | 11 (11) | 10 (10) | 3 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (9) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 8 (8) | 13 (13) | 3 (3) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 55 (56) | 104 (105) | 6 (6) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 28 (29) | 51 (51) | 2 (2) | 7 (7)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 6 (7) | 6 (6) | 2 (2) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (3) | 3 (5) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 13 (17) | 25 (27) | 6 (6) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 8 (9) | 11 (11) | 5 (5) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 11 (12) | 7 (7) | 0 (0) | 2 (2)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 66 (68) | 77 (79) | 3 (3) | 6 (7)
Rib fracture (Injury, poisoning and procedural complications) | 7 (9) | 10 (10) | 2 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Sternal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) | 3 (3) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 12 (13) | 23 (28) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 13 (13) | 22 (22) | 3 (3) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 15 (17) | 28 (28) | 3 (3) | 3 (4)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (7) | 1 (1) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cortisol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Grip strength decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Residual urine volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 13 (13) | 7 (7) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 10 (10) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 (8) | 9 (9) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperosmolar state (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (9) | 6 (6) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 14 (15) | 4 (4) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 2 (2) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 12 (13) | 8 (10) | 2 (2) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 22 (22) | 1 (1) | 1 (1)
Bone loss (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 12 (14) | 10 (11) | 1 (1) | 0 (0)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (10) | 1 (1) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint adhesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 0 (0) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Morphoea (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 135 (154) | 115 (132) | 12 (12) | 12 (13)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 4 (4) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 18 (18) | 11 (12) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 15 (15) | 17 (17) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ulnocarpal abutment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 7 (8) | 2 (2) | 1 (1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 79 (93) | 71 (87) | 9 (10) | 8 (9)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 (33) | 32 (32) | 4 (4) | 9 (9)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Clear cell endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (23) | 17 (17) | 4 (4) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicle centre lymphoma, follicular grade I, II, III stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5) | 3 (3) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (1) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 23 (24) | 4 (4) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metaplastic breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed adenoneuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ovarian epithelial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 9 (9) | 3 (3) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (5) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 12 (12) | 4 (5) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (20) | 10 (10) | 3 (3) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apallic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 9 (11) | 5 (5) | 2 (2) | 2 (2)
Cerebellar infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 9 (9) | 2 (2) | 3 (3)
Cerebral infarction (Nervous system disorders) | 31 (32) | 18 (18) | 1 (1) | 5 (5)
Cerebral ischaemia (Nervous system disorders) | 5 (5) | 8 (9) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 68 (68) | 42 (43) | 8 (8) | 4 (4)
Cerebrovascular disorder (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Cerebrovascular insufficiency (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (10) | 7 (7) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslalia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 6 (7) | 2 (2) | 0 (0) | 1 (1)
Frontotemporal dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 6 (6) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 39 (40) | 40 (41) | 21 (22) | 7 (7)
Lacunar infarction (Nervous system disorders) | 4 (4) | 8 (9) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 6 (6) | 8 (8) | 4 (4) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningorrhagia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Parkinsonism (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 6 (7) | 2 (3) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 5 (5) | 1 (1) | 3 (3)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Slow speech (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 31 (33) | 20 (20) | 4 (5) | 4 (4)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 31 (33) | 35 (38) | 2 (2) | 3 (3)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compulsive hoarding (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 10 (10) | 10 (10) | 0 (0) | 1 (1)
Dysphemia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychogenic pain disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 6 (6) | 1 (1) | 2 (2)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 5 (5) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 10 (10) | 2 (2) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleroderma renal crisis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urethral caruncle (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anisomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 7 (7) | 2 (2) | 1 (1) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrometra (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 12 (12) | 5 (5) | 1 (1) | 3 (3)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Vaginal polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 14 (15) | 13 (14) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 7 (7) | 10 (10) | 1 (1) | 1 (1)
Vulval leukoplakia (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vulvar dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 9 (9) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 17 (20) | 2 (2) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 34 (43) | 36 (44) | 9 (11) | 5 (6)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 2 (2) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal pouch (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 8 (8) | 3 (3) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 4 (4) | 0 (0)
Pulmonary arteriopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 28 (30) | 7 (7) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Pulmonary ossification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 9 (9) | 1 (1) | 1 (1)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus polyp degeneration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Atrophoderma of Pasini and Pierini (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 3 (3) | 2 (2)
Skin wrinkling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Immobile (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 8 (9) | 4 (4) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic disorder (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 17 (19) | 9 (9) | 1 (1) | 3 (3)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Iliac artery embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extremity necrosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 31 (34) | 37 (39) | 2 (2) | 4 (4)
Hypertensive crisis (Vascular disorders) | 10 (12) | 20 (21) | 4 (4) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 3 (3) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infarction (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 4 (4) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (8) | 5 (6) | 3 (3) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Peripheral circulatory failure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 8 (8) | 3 (3) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ciliary body disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical leukoplakia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study + First Extension: Odanacatib 50 mg OW (N=8043) | Base Study + First Extension: Placebo (N=8028) | Second Extension: Odanacatib 50 mg OW (N=3144) | Second Extension: Odanacatib 50 mg OW (Placebo) (N=2309)
Anaemia (Blood and lymphatic system disorders) | 477 (552) | 500 (583) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 488 (638) | 492 (652) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 492 (547) | 504 (552) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 589 (726) | 504 (608) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 450 (591) | 459 (611) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 495 (610) | 443 (564) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 957 (1396) | 938 (1365) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 644 (962) | 596 (913) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1724 (2911) | 1699 (2821) | 311 (393) | 209 (271)
Accidental overdose (Injury, poisoning and procedural complications) | 476 (761) | 499 (736) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 386 (500) | 422 (568) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1221 (1588) | 1151 (1533) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1194 (1473) | 1136 (1394) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 518 (589) | 461 (537) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 785 (980) | 741 (910) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 751 (923) | 671 (797) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 492 (574) | 483 (565) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 471 (553) | 466 (544) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1104 (1263) | 1084 (1278) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to an observed increase in risk of stroke in Protocol MK-0822-018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.